

### PM1183-A-019-20

An Open-Label, Multicenter Study to Assess the Potential Effects of Bosentan (a Moderate CYP3A4 Inducer) on the Pharmacokinetics of Lurbinectedin in Patients with Advanced Solid Tumors

#### STATISTICAL ANALYSIS PLAN

INVESTIGATIONAL MEDICINAL PRODUCTS: Lurbinectedin (Zepzelca®), and

Bosentan.

**Protocol No.:** PM1183-A-19-20 **EudraCT No.:** 2020-002595-12 **NCT Code:** NCT05072106

Version: v2.0

Date: 18-MAR-2022

## TABLE OF CONTENTS

| 1 | STUI | DY RATIONALE | 6 |
|---|---|---|---|
| 2 | OVE: | RALL STUDY DESIGN | 6 |
| 3 | PATI | ENTS EVALUABILITY CRITERIA | 9 |
| 4 | OBJE | CTIVES AND ENDPOINTS | . 10 |
| | | bjectives | |
| | 4.1.1 | Primary Objective | . 10 |
| | 4.1.2 | Secondary Objective | . 10 |
| | 4.2 E | ndpoints | . 10 |
| | 4.2.1 | Primary Endpoint | . 10 |
| | | Secondary Endpoint | |
| 5 | | PLE CONSIDERATIONS | |
| | | andomization | |
| | | ample Size | |
| 6 | | TISTICAL METHODOLOGY | |
| | | oxicity and Adverse Events | |
| | | linical Laboratory Evaluation | . 12 |
| | | hysical Examination, Vital signs, Left Ventricular Ejection Fraction and | |
| | | ardiogram Findings | |
| | | eaths and other Serious Adverse Events | |
| 7 | | ER ANALYSES | |
| | 7.1 B | aseline and Demographics | . 13 |
| | | atient Disposition and Treatment/Study Discontinuation | |
| | | rotocol Deviations | |
| | | reatment Administration | |
| | | ubsequent Therapies | |
| | | ubgroup Analyses | |
| | | harmacogenetics Analyses | |
| | | ecimal places | |
| | | mputation in Incomplete Dates | |
| | 7.10 | Variable Unit Standardization | |
| | 7.11 | Decimal Places, Missing Values and Allowed Assessment Windows | |
| 0 | 7.12 | Identification of Fixed or Random Effects Models | |
| 8 | | TISTICAL SOFTWARE | |
| 9 | | RENCES | |
| 1( | | ENDIX I: PATIENTS DISPOSITION | |
| | 10.1 | General Characteristics | |
| | 10.1. | 1 | |
| | 10.1.2 | | |
| | 10.1.3 | | |
| | 10.2 | Patient Characteristics | |
| | 10.2. | $\mathcal{E}_{-1}$ | |
| | 10.2.2<br>10.2.3 | J | |
| | 10.2.4 | J | |
| | | I J | |
| | 10.2.3 | , | |
| | 10.2.0 | | |
| | 10.2. | Biochemical Evaluation at Baseline | . 49 |

| | 10.2.8 | Coagulation Evaluation at Baseline | 30 |
|-----|---------|------------------------------------------|----|
| | 10.2.9 | Signs and Symptoms at Baseline | 30 |
| | 10.2.10 | Concomitant Medication at Baseline | 31 |
| 11 | APPEN | DIX II: SAFETY ANALYSIS | 32 |
| 1 1 | 1.1 | Extent of exposure | 32 |
| | 11.1.1 | Treatment Administration | 32 |
| | 11.1.2 | Cycle Delays | 33 |
| | 11.1.3 | Dose Reductions | 34 |
| | 11.1.4 | Any Other Dose Modifications | 34 |
| 1 | 1.2 | Adverse Events (AEs) | 35 |
| | 11.2.1 | Display of Adverse Events | 35 |
| 1 1 | 1.3 | Serious Adverse Events and Deaths | 38 |
| | 11.3.1 | Serious Adverse Events | 38 |
| | 11.3.2 | Deaths | 39 |
| 1 | 1.4 | Clinical Laboratory Evaluation | 40 |
| | 11.4.1 | Hematological Abnormalities | 40 |
| | 11.4.2 | Biochemical Abnormalities | 41 |
| | 11.4.3 | Laboratory Values Over Treatment | 42 |
| 1 | 1.5 | Linear Mixed-effects Model | 44 |
| 11 | 1.6 | Physical Findings, ECOG PS, LVEF and ECG | 44 |
| | 11.6.1 | Physical Findings and ECOG PS | |
| | 11.6.2 | LVEF and ECG | |
| 1 | 1.7 | Concomitant Therapies | 45 |
| | 11.7.1 | Concomitant Medication during the Study | 45 |
| | 11.7.2 | Further Antitumor Therapies | |
| 12 | APPEN | DIX III: EFFICACY ANALYSIS | 46 |
| 13 | APPEN | DIX IV: DB Listings | 47 |
| 14 | APPEN | DIX V: BIMO Listings | 51 |
| 15 | APPEN | DIX VI: ICH Listings | 53 |
| 16 | | DIX VI: VERSION HISTORY | |
| 16 | 5.1 | History of Changes | 54 |

#### ABBREVIATIONS AND GLOSSARY

**AE(s)** Adverse Event(s)

ALT Alanine Aminotransferase AP Alkaline Phosphatase AST Aspartate Aminotransferas

AST Aspartate Aminotransferase

ATC Anatomical Therapeutic Chemical

**AUC** Area Under the Concentration-time Curve

**BIMO** Bioresearch Monitoring

**BOS** Bosentan

BSA Body Surface Area
CI Confidence Interval

Cl Clearance

C<sub>max</sub> Maximum Plasma Concentration

**CPK** Creatine Phosphokinase

**CPK-MB** Creatine Phosphokinase Isoenzyme MB

CrCl Creatinine Clearance
CRF Case Report Form
CRP C-reactive Protein
CV Coefficient of Variation
CYP Cytochrome P450

**D** Dav

**DL** Dose Level

DSBs Double-strand Breaks
ECG Electrocardiogram
ECHO Echocardiogram

**ECOG PS** Eastern Cooperative Oncology Group Performance Status

**EDC** Electronic Data Capture

**EOT** End of treatment

**FDA** Food and Drug Administration

GCP Good Clinical Practice
GGT Gamma-glutamyltransferase

IC50 Half Maximal Inhibitory Concentration ICH International Conference on Harmonization

**INR** International Normalized Ratio

**i.v.** Intravenous

L Liter

**LDH** Lactate Dehydrogenase

**LRB** Lurbinectedin

**LVEF** Left Ventricular Ejection Fraction

MedDRA Medical Dictionary for Regulatory Activities

Mg Milligram mL Milliliter

MUGA Multiple-gated Acquisition Scan

NA Not Applicable

NCI-CTCAE National Cancer Institute Common Toxicity Criteria

PD Progressive Disease
PGt Pharmacogenetic
PK Pharmacokinetics
PS Performance Status

PT Preferred Term
q3wk Every Three Weeks
RBC Red Blood Cells

**RT** Reference-Test Sequence

**RTSM** Randomization and Trial Supply Management

SAE(s)Serious Adverse Event(s)SAPStatistical Analysis PlanSCLCSmall Cell Lung Cancer

**SmPC** Summary of Product Characteristics

SOC System Organ Class
 Std. Standard Deviation
 T<sub>1/2</sub> Terminal Half-life

TR Test-Reference Sequence ULN Upper Limit of Normal

Vss Volume of Distribution at Steady State

**WBC** White Blood Cells

WHO World Health Organization

wk Week(s)

#### 1 STUDY RATIONALE

Lurbinectedin is a novel synthetic tetrahydroisoquinoline structurally related to ecteinascidins.

Lurbinectedin is a new chemical entity that binds the DNA leading to the formation of DNA double-strand breaks (DSBs). The binding to DNA is likely occurring in the minor groove region and induces apoptosis and delayed progression through the cellular phase S/G2. Lurbinectedin also induces the specific degradation of transcribing RNA Pol II in several human tumor cell lines.

In vitro, lurbinectedin demonstrated cytotoxic effects against a broad selection of tumor types with half maximal inhibitory concentration (IC50) values in the range of 1-10 nM. Although selectivity was also seen, a clustering of sensitive tumors has not been identified. Lurbinectedin also exhibited antitumor activity against different murine models of xenografted human-derived tumor types. Lurbinectedin has been tested as a single agent or in combination with different drugs in solid tumors; while antitumor activity in hematological tumors was deemed negligible, lurbinectedin has shown activity in different solid tumors; some of the most responsive tumor types were breast, small cell lung cancer (SCLC), ovarian and endometrial cancer.

Based on current clinical data, the toxicity of lurbinectedin is predictable, reversible and manageable. The most relevant toxicity is reversible myelosuppression with a nadir occurring in the middle of the second week after Day 1 infusion in an every-three-week cycle; overall, the incidence of febrile neutropenia is below 20% in all ongoing Phase II trials.

Lurbinectedin is extensively metabolized by the cytochrome P450 enzymes, primarily CYP3A4. Thus, potent inducers or inhibitors of this enzyme may alter the plasma concentrations of lurbinectedin. This study is designed to examine the pharmacokinetics (PK) and safety of lurbinectedin when co-administered with bosentan, a moderate CYP3A4 inducer, in comparison with lurbinectedin alone. The results of this study may be used to support future clinical studies in patients and prescribing information in future labeling.

A full rationale for the study may be found in the appropriate sections of the study's clinical protocol.

#### 2 OVERALL STUDY DESIGN

This is a prospective, open-label, two-way crossover, phase Ib drug-drug interaction study in patients with advanced solid tumors.

The study will include a pre-treatment (screening) phase (within 14 days before the first lurbinectedin or bosentan administration) followed by a treatment phase consisting of two lurbinectedin cycles, one cycle in combination with bosentan and one cycle of lurbinectedin as single agent (in different order depending on the study sequence), and one additional third cycle of lurbinectedin as a single agent for patients who meet the continuation criteria and obtain a clinical benefit after the first two cycles, and then follow-up of adverse events if any.

Patients who meet the continuation criteria and obtain a clinical benefit according to the Investigator's criteria will have the opportunity to continue treatment under a Compassionate Use Agreement after the completion of the optional third study cycle.

Patients will be treated as outpatients. At the discretion of the Investigator, patients may be admitted to the study center on Day -1 or Day 1 and monitored, at least, until completion of the Day 1 PK blood sample collections.

Patients will receive a maximum of three cycles: two consecutive cycles of lurbinectedin, one cycle with and one cycle without bosentan co-administration (in different order depending on the study Sequence 1 or Sequence 2 of treatment), followed by a third cycle with lurbinectedin alone (this last optional for patients with clinical benefit). Lurbinectedin will be administered as a 1-hour (-5/+20 min) i.v. infusion every three weeks (q3wk) via a central or peripheral vein.

In the co-administration cycles, bosentan will be administered orally twice daily in the morning and evening during the prior five consecutive days, self-administered at home from Day -5 to Day -1 (i.e., five days before lurbinectedin infusion), and once daily on Day 1 (i.e., the day of lurbinectedin infusion), following recommendations at the Summary of Product Characteristics (SmPC). On Day 1 (i.e., the day of lurbinectedin infusion), bosentan will be given immediately prior to starting the lurbinectedin infusion. In fact, bosentan should be administered after obtaining the bosentan PK sample #1 and before the start of lurbinectedin infusion (-15 min to -1 min).

In case of lurbinectedin delay ( $\leq 2$  days), bosentan could be administered twice daily during a maximum of seven consecutive days before lurbinectedin infusion, and supplied at the study center once daily on Day 1 (before lurbinectedin infusion).

All patients will receive a maximum of three cycles: two consecutive cycles of lurbinectedin, one cycle with and one cycle without bosentan co-administration (in different order depending on the study Sequence 1 or Sequence 2 of treatment), followed by a third cycle with lurbinectedin alone (this last optional for patients with clinical benefit).

Patients will be randomized in a 1:1 ratio to Sequence 1 (TR: Test- Reference; lurbinectedin + bosentan in Cycle 1) or Sequence 2 (RT: Reference-Test; lurbinectedin + bosentan in Cycle 2). Lurbinectedin will be administered as a 1-hour (-5/+20 min) intravenous (i.v.) infusion q3wk via a central or peripheral vein. The dose of lurbinectedin will be 3.2 mg/m² for all patients when administered with and without bosentan. If toxicity occurs, the appropriate intra-patient dose level (DL) reductions will be implemented in the subsequent cycle.



The enrollment of the patients will be simultaneous. However, if once the first three patients enrolled have completed Cycle 1 and Cycle 2, total lurbinectedin exposure does not allow an adequate PK assessment and if no unacceptable or life-threatening toxicities have occurred, the dose of lurbinectedin to be co-administered with bosentan in the remaining five patients can be adjusted accordingly.

This decision will be made by the Sponsor and the study Investigators. Therefore, the planned dose of lurbinectedin, when given with bosentan for the remaining five patients, will be based on the acceptability of the PK and safety results from the first three patients. If the initial three patients do not experience adverse events (AEs) which might require a dose-reduction, the dose of lurbinectedin may still be adjusted (based on the assumption of dose-proportional pharmacokinetics) to produce plasma lurbinectedin area under the curve (AUC) values that are comparable to those when lurbinectedin is given in the absence of bosentan. However, if toxicity occurs in the initial three patients, the appropriate dose-reduction of lurbinectedin will be implemented in the remaining five patients accordingly.

Patients will receive lurbinectedin until disease progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest, and for a maximum of three cycles. Treatment with lurbinectedin outside this study could be continued under a Compassionate Use Agreement after the completion of the optional third study cycle.

All patients will be randomly assigned to the corresponding sequences:

- Sequence 1 (TR):
- o Cycle 1: Bosentan + lurbinectedin
- o Cycle 2: Lurbinectedin alone
- Cycle 3: Lurbinectedin alone (optional)
- Sequence 2 (RT):
- o Cycle 1: Lurbinectedin alone
- o Cycle 2: Bosentan + lurbinectedin
- Cycle 3: Lurbinectedin alone (optional)

Lurbinectedin will be administered to eight evaluable patients and for a maximum of three cycles, while considered to be on the patient's best interest or until progressive disease (PD), unacceptable toxicity, intercurrent illness of sufficient magnitude to preclude safe continuation of the study, patient's refusal and/or non-compliance with study requirements, a protocol deviation with an effect on the risk/benefit ratio of the clinical study or any other reason at the physician's judgment that precludes lurbinectedin continuation.

If the patient responds to treatment after the first two cycles according to Investigator criteria for clinical benefit, treatment with lurbinectedin may continue outside this study under a Compassionate Use Agreement at the same dose based on Investigator's decision and upon agreement with the Sponsor. Then, the treating center must request authorization to the relevant Health Authorities and notify the Sponsor in due time. In order to avoid a treatment discontinuation, during the Compassionate Use Agreement authorization an additional third cycle with lurbinectedin is allowed.

All AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5. Treatment delays, dose reduction requirements and reasons for treatment discontinuation will be monitored throughout the study. The safety profile of patients will be monitored throughout the treatment and up to 31 days (±10 days) after the last lurbinectedin infusion (end of treatment, EOT), until the patient starts a new antitumor therapy or until the date of death, whichever occurs first. Any treatment-emergent AEs will be followed until recovery to at least grade 1 or stabilization of symptoms or until the start of a new antitumor therapy, until the continuation of treatment outside this study under a Compassionate Use Agreement or death, whichever occurs first. After treatment discontinuation, patients will be followed until resolution or stabilization of all toxicities, if any.

Patients will be evaluated at scheduled visits on three study periods: pre-treatment (screening), treatment (one cycle of lurbinectedin in combination with bosentan and two as a single agent and the third cycle optional) and follow-up of adverse events if any.

#### 3 PATIENTS EVALUABILITY CRITERIA

Patients must fulfill all the inclusion/exclusion criteria to be enrolled in the study.

The study will include the following analysis population set definitions:

- The <u>enrolled population</u> is defined as all patients recorded in the database who have been included in the trial and randomized, regardless of whether they have received the study drug or not. Screening failure patients will not be considered as part of this population.
- The <u>PK population</u> will include all patients who have provided sufficient and interpretable PK parameters to calculate the non-compartmental PK parameters. Evaluable patients should have received the first two complete cycles regardless dose delays or reductions.
- The <u>safety population</u> will include all patients who received at least one dose of lurbinectedin. Patients who have received at least one dose of bosentan but who did not receive any dose of lurbinectedin will be excluded from the safety population and will be performed separately by narratives. The safety population will be used for all safety evaluations.

#### 4 OBJECTIVES AND ENDPOINTS

#### 4.1 Objectives

This clinical pharmacology study is designed to assess the impact of bosentan co-administration on lurbinectedin PK parameters administered alone.

#### 4.1.1 Primary Objective

• To assess the effect of bosentan on lurbinectedin total plasma exposure in patients with advanced solid tumors.

#### 4.1.2 Secondary Objective

- To assess the effect of bosentan on lurbinectedin unbound plasma exposure.
- To assess the effect of bosentan on lurbinectedin major metabolites (i.e., M1 and M4).
- To assess the effect of bosentan on the safety profile of lurbinectedin.
- To collect and store a blood sample for germline DNA extraction for future pharmacogenetic (PGt) analysis of variations on genes that may influence exposure and response (i.e., disposition, metabolism and safety) to lurbinectedin.

#### 4.2 Endpoints

#### 4.2.1 Primary Endpoint

• Plasma dose-normalized  $C_{max}$  and  $AUC_{0-\infty}$  of lurbinectedin will be compared between Cycle 1 and Cycle 2. Pharmacokinetic analyses will be evaluated in plasma by standard non-compartmental methods, or population methods, if necessary.

#### 4.2.2 Secondary Endpoint

- Differences in dose-normalized total AUC<sub>0-t</sub> and C<sub>max</sub> and in Cl, Volume of Distribution at Steady State (V<sub>ss</sub>) and T<sub>1/2</sub> of lurbinectedin between Cycle 1 and Cycle 2 will be explored.
- Differences in dose-normalized unbound  $AUC_{u,0-\infty}$ ,  $AUC_{u,0-t}$  and  $C_{u,max}$  and in  $CL_u$ ,  $V_{ss,u}$  and  $T_{1/2,u}$  of lurbinectedin between Cycle 1 and Cycle 2 will be explored.
- Differences in ratios between total AUC<sub>0-∞</sub>, AUC<sub>0-t</sub> and C<sub>max</sub>, of main lurbinectedin metabolites relative to parent drug between Cycle 1 and Cycle 2 will be explored. Additional PK parameters will be calculated if deemed appropriate.
- Treatment safety, including AEs, serious adverse events (SAEs) and laboratory abnormalities will be graded according to the NCI-CTCAE v.5. Additionally, treatment compliance, in particular dose reductions requirements and/or treatment delays due to AEs, and reasons for treatment discontinuation will also be described. Patients will be evaluable for safety if they have received at least one partial or complete infusion of lurbinectedin.

• The presence or absence of pharmacogenetic (PGt) polymorphisms in genes relevant for lurbinectedin disposition (distribution, metabolism and excretion) from a single blood sample collected (only if written IC given) at any time during the trial (but preferably at the same time as the pre-treatments PK sample on Day 1 of Cycle 1), which will be stored to explain individual variability in main PK parameters in future analyses.

#### 5 SAMPLE CONSIDERATIONS

#### 5.1 Randomization

A block randomization (1:1 ratio) will be performed to avoid bias in the assignment of patients to treatment sequence group, to increase the likelihood that known and unknown subject attributes (e.g., demographic and baseline characteristics) are evenly balanced across treatment sequence groups, and to enhance the validity of statistical comparisons across treatment sequence groups.

At least eight patients are expected to complete all study procedures, including the collection of sufficient and interpretable PK assessments. Although at least eight patients will be enrolled in this study; it is estimated that complete data from eight patients will be sufficient to estimate the drug-drug interaction of bosentan on the PK of lurbinectedin.

Randomization will apply for all patients.

Patients must be replaced if they are not evaluable for the assessment of the primary endpoint (e.g., if they have not sufficient and interpretable PK parameters).

Randomization will be implemented in Medidata Rave RTSM. A randomization list will be generated to randomly allocate patients to Sequence 1 (TR: Test- Reference; lurbinectedin + bosentan in Cycle 1) or Sequence 2 (RT: Reference-Test; lurbinectedin + bosentan in Cycle 2). Additional randomization lists will be generated in case non-evaluable patients need to be replaced. Variable block sizes and allocation ratios will be used depending on the number of patients to be replaced in each case scenario in order to complete both sequence treatment groups while keeping balance across them. In order to achieve reproducible results, the seed used in the generation of each randomization list will be saved.

#### 5.2 Sample Size

This study was designed to assess the potential effects of bosentan on the PK of lurbinectedin in patients with advanced malignancies. The 90% confidence interval (CI) will be used to help with the interpretation of the results. A sample size of eight patients was based on feasibility and clinical considerations. Based on previous studies, the intra-subject coefficient of variation (CV) of lurbinectedin PK parameters is estimated to be more than 30%. The precision (half-width) of the 90% CI for [(lurbinectedin + bosentan) / lurbinectedin alone] comparison on the log-scale will extend 0.389 from the observed differences in means, assuming that the intra-subject CV around 40%. This half-width corresponds to a 90% CI in the range of 70% and 147% assuming the ratio of the means equal to unity for each PK parameter. This 90% CI will be used to help with the interpretation of the results.

#### 6 STATISTICAL METHODOLOGY

The PK definitions and analysis plan will be described by the Clinical Pharmacology department in a separate document. The present Statistical Analysis Plan (SAP) is focused on the statistical methodology for safety.

Safety analyses will consider treatment emergent AEs and SAEs, according to their relationship with study treatment, as well as analytical results, deaths and the reasons for treatment discontinuations, delays and/or dose reductions.

All AEs and SAEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

Descriptive statistics will be used to characterize the profiles of drug-related AEs, drug-related deaths, SAEs, clinical laboratory data, drug-related delays and/or treatment discontinuations. Tables will be displayed by sequence and treatment (Sequence 1 [TR] vs. Sequence 2 [RT]) and treatment group (Test [lurbinectedin administered in combination with bosentan] vs. Reference [lurbinectedin alone]).

#### 6.1 Toxicity and Adverse Events

The toxicity evaluation will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v.5).

Summary of overall AEs will be done by system organ class (SOC) and preferred term (PT), by severity (worst toxicity grade) and by relationship to the study drug (any of them or both). Tables will be sorted by category of events using SOC and PT.

#### 6.2 Clinical Laboratory Evaluation

Laboratory results will be classified according to the NCI-CTCAE v.5.

All laboratory visits reported as "End of treatment" visit will be mapped to the last cycle visit for each patient. Worst grade per patient and per cycle for applicable values during treatment will be shown.

The following hematological values will be displayed: hemoglobin, erythrocytes (RBC), white blood cells count (WBC), neutrophils, lymphocytes, monocytes, hematocrit and platelets count.

For the analysis by sequence, overall cross tabulation will be presented for the worst grade during treatment vs. the baseline toxicity grading of anemia, lymphopenia, neutropenia, leukopenia and thrombocytopenia.

If a grade  $\geq 3$  neutropenia or thrombocytopenia occurs during a treatment cycle, the first day it reaches grade 3 or 4 (counting from the start of the cycle) and the duration of the abnormality (i.e., until recovery to grade  $\leq 2$ ) will be tabulated. The information will be shown by means of median and range.

The following biochemical and coagulation values will be displayed: aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline Phosphatase, lactate dehydrogenase (LDH), creatinine, creatinine clearance, glucose, creatine phosphokinase (CPK), CPK-MB fraction, gamma glutamyltransferase (GGT), total bilirubin, direct bilirubin, serum electrolytes (Na+, K+, Mg++), total calcium, total proteins, albumin, Creactive protein count (CRP) and the international normalized ratio (INR).

If a grade  $\geq 3$  AST or ALT increase occurs during a treatment cycle, both the day it peaked and the duration of the abnormality will be tabulated. The information will be shown by means of median and range.

Overall cross tabulation will be presented for the worst grade during treatment vs. the baseline toxicity grading of biochemical abnormalities.

# 6.3 Physical Examination, Vital signs, Left Ventricular Ejection Fraction and Electrocardiogram Findings

Tables summarizing the performance status (PS), height, body weight and body surface area (BSA), vital signs, left ventricular ejection fraction (LVEF) at baseline and during the treatment will be prepared.

If appropriate, changes in the ECOG PS and body weight of each patient during the treatment compared with baseline will also be done.

Cardiac rhythm will be done in triplicate and identified ECG intervals of at least 30 seconds of duration, PR interval and QT interval (raw and corrected by HR using Bazett's formula). Mean of all ECGs collected on each time point will be used for analysis.

#### 6.4 Deaths and other Serious Adverse Events

Deaths and other serious adverse events (SAEs) will be tabulated following the same pattern than AEs. In addition, all deaths within 60 days from the first dose of treatment or within 30 days from the last dose of treatment will be listed.

#### 7 OTHER ANALYSES

Descriptive statistics (mean, median, standard deviation, range of value, frequencies and percentages) will be used to summarize the data. Counts and percentages will be used for categorical variables, and summary tables will be used for continuous variables.

#### 7.1 Baseline and Demographics

Descriptive statistics will be used to summarize the patients' baseline characteristics

Baseline data such as demographics, cancer history, prior therapy, prior relevant history, signs and symptoms, ECG, LVEF, physical examination, vital signs, laboratory values and concomitant medication, coded according to the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system, will be described following standard tables (detailed in Section10, Appendix I).

Age, baseline weight, height and BSA values will be summarized descriptively. Age categories, sex, race and baseline ECOG PS will be summarized with frequency counts.

For the cancer history, times from initial diagnosis, metastatic disease, from locally advanced disease and from last progression before the study entry will be summarized. These time calculations will be shown in months and summarized descriptively. Histology and characteristics of the disease at study entry will be tabulated.

Previous relevant medical history (other than cancer) will be listed.

A frequency tabulation of the number of patients with the different types of previous surgery, radiotherapy or therapy will be given.

Signs and symptoms will be displayed by tabulation of frequencies according to NCI-CTCAE v.5 toxicity grades. Signs and symptoms will be listed.

In case of pre-treatment characteristics with multiple measurements per subject before the start of treatment (e.g. laboratory assessments or vital signs), the last value prior to or on the first day of treatment will be considered the baseline measurement.

#### 7.2 Patient Disposition and Treatment/Study Discontinuation

The number of patients included and treated in the study will be shown. Also, accrual by center and the main dates of the study will be displayed. Reasons for treatment discontinuation and for study discontinuation will be tabulated.

#### 7.3 Protocol Deviations

Analysis of inclusion/exclusion criteria deviations, retreatment restrictions, concomitant medication and clinically relevant discontinuations, among others, will be done as described in Appendix I.

#### 7.4 Treatment Administration

Exposure to treatment will be described by treatment group.

Total cumulative dose, time on treatment, dose intensity and relative dose intensity, administration delay and dose reductions/omissions will be described following standard tables (detailed in Section 11, Appendix II). The reported cycle information on the case report form (CRF) pages will be used for the analysis.

Time on treatment, expressed in weeks, is defined as the last administration date of lurbinectedin minus the first administration date plus 31 days, except if the patient dies or starts a new antitumor therapy within 31 days from the last administration date, in which case the time on treatment will be the date of death or the start date of the new antitumor therapy minus the date of the first administration of the study treatment.

Total cumulative dose by drug, expressed in mg for both lurbinectedin and bosentan, is the sum of all the product doses received during the study, including the dose received in the last cycle.

For lurbinectedin, intended dose intensity is the planned dose per cycle divided by the planned number of weeks by cycle.

Absolute dose intensity is the actual cumulative dose divided by the number of weeks of treatment. As a convention, for this calculation, the duration of the last cycle will be the predefined cycle length (e.g, 21 days). Relative dose intensity (%) is the ratio of absolute dose intensity divided by the intended dose intensity.

The items « Infusion delayed: yes/no» and « Dose reduced: yes/no» present on the treatment exposure CRF pages will be used to calculate delays and dose reductions, respectively. For cycles considered as delayed by the Investigator, the length of the delay will be calculated as:

Duration of cycle delay: Date of the current drug administration – Date of the previous drug administration – the predefined cycle length (i.e., 21 days).

If the number of delays or dose reductions are very low, tables will not be presented and only listings will be shown.

#### 7.5 Subsequent Therapies

A listing of subsequent therapies received after treatment discontinuation will be shown by total and treatment sequence group.

#### 7.6 Subgroup Analyses

Safety analysis will be done by sequence (Sequence 1 [TR] vs Sequence 2 [RT]) and treatment group (Test [lurbinectedin administered in combination with bosentan] vs Reference [lurbinectedin alone]). Additional groups could be done (such a dose level in case dose of lurbinectedin was adjusted) if required, and a sequential number will be added at the end of the table number to differentiate them within each section.

No other subgroup analysis is planned.

#### 7.7 Pharmacogenetics Analyses

The analysis will be detailed and reported in a separate document.

#### 7.8 Decimal places

By default, all results will be rounded to one decimal, except when variables are integers; in that case, they will be reported without decimals, (e.g. age in years or number of sites).

### 7.9 Imputation in Incomplete Dates

The dates of certain historical or current clinical activities are key component for statistical analysis. An incomplete date results from a missing day, month or year; in that case, the missing figure can be imputed allowing for the calculation of variables, such duration and time to certain event. However, when all of them, day, month and year, are missing no imputation will be done.

#### Before randomization/treatment start date

All variables needed to summarize for example prior information (e.g. first diagnosis date) where partial information is available will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month is also unknown then the imputed date will 1/July. This assumption will be valid if the imputed date is earlier than the randomization date; otherwise, the imputed date will be the first day of the month of the randomization date (i.e. 01/Randomization month date/year).

#### Between treatment start and end of treatment

All date variables during treatment where information is needed and is not fully available, for example adverse events or concomitant medications, will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month and/or year is also unknown then the imputed date will be 1/January (this assumption will be valid if the imputed date is not earlier than the treatment start date; otherwise, the imputed date will be the treatment start date).

#### After end of treatment

A conservative approach for the variables collecting information after end of treatment where partial information is available (e.g., follow-up AEs) will be imputed by means of SAS programming. The following rules will be implemented: if the day of a date is unknown then the imputed day will be 1; if the month is also unknown, then the imputed date will be 1/July. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise, the imputed date will be the last study drug administration date plus 1 day.

#### 7.10 Variable Unit Standardization

Variables reported with different units will be homogenized to standardized variables following the International System of Units (e.g. laboratory tests, biometrical assessments...) unless otherwise specified in the following sections.

#### 7.11 Decimal Places, Missing Values and Allowed Assessment Windows

By default, all numeric results will be rounded to one decimal place, except when variables are integer, which will be reported without decimals (e.g., age in years, number of sites, etc.). Four decimals will be used for p-values.

Missing values will not be included in the calculation of percentages. Assessment windows as specified in the clinical protocol will be respected.

#### 7.12 Identification of Fixed or Random Effects Models

Not applicable (NA).

#### 8 STATISTICAL SOFTWARE

Medidata Rave<sup>®</sup> EDC will be used for data entry and clinical data management.

Medidata Rave® RTSM will be used for permuted block randomization design and management.

SAS® v.9.4 or superior will be used for all statistical analysis outputs.

#### 9 REFERENCES

• Food and Drug Administration (FDA).2001. Guidance for Industry. Statistical approaches to establishing bioequivalence.

#### 10 APPENDIX I: PATIENTS DISPOSITION

#### 10.1 General Characteristics

The general characteristics analysis will be carried out on the enrolled population.

#### 10.1.1 Patient Disposition

Main characteristics concerning inclusion in the study, withdrawal from the study and protocol deviations will be displayed in this section.

Table 10.1.1.1 Patient accrual by institution

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

Institution 1

Institution 2

Total

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### Table 10.1.1.2 Disposition of patients

Relevant study dates

Date of first consent

Date of first dose/first patient

Date of last consent

Date of first dose/last patient

Date of last dose

Date of last follow up\*

(\*) Last follow up date, examination date or procedure before study closure.

Table 10.1.1.3 Number of patients evaluable for analysis

| _ | S1 (TR) | | S2 (RT) | | Total | |
|---|---------|---|---------|---|-------|---|
| | N | % | N | % | N | % |

Evaluable for Safety

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 10.1.1.4 Non-evaluable patients

| Not Evaluable for | Sequence | Subject | Reason(s) |
|-------------------|----------|---------|-----------|
| Safety | | | |
| PK | | | |

### 10.1.2 Treatment Discontinuations

| OD 11 1 | Λ 1 | A 1 | OD 4 | 1. | |
|----------|------|---------|------------|-------|-------------|
| Lable L | () [ | · / I | Treatment | dieco | ntiniiation |
| I abic I | υ. ι | . 4 . 1 | 11 Cauncin | uisco | mmuanon |

| | | | S1 (TR) | | S2 (RT) | | Total | |
|---|---|---|---|---|---|---|---|---|
| | | | N | % | N | % | N | % |
| Protocol Treatme | ent Completed | | | | | | | |
| Patient moved to | Compassionate | Use | | | | | | |
| Progressive disea | ise | | | | | | | |
| Adverse Events | | | | | | | | |
| Patient refusal to | treatment | | | | | | | |
| Investigator's dec | cision | | | | | | | |
| Death | | | | | | | | |
| Other | | | | | | | | |
| Total | | | | | | | | |
| Listing 10.1.2.2 | | | | | | | l.: ( | Saniana Enand |
| Listing 10.1.2.2<br>Sequence | 2 Treatment di<br>Subject | scontinuation d<br>AE reported | ue to rela Preferre | | verse Event<br>Grade | s<br>Relations | hip S | Serious Event |
| Sequence | Subject | AE reported | | | | | hip S | Serious Event |
| Sequence | Subject | AE reported | | | | | hip S | Serious Event |
| Sequence Notes: † Related of Listing 10.1.2.3 | Subject<br>or unknown rela | AE reported | Preferre | d term | Grade | Relations) | | Serious Event |
| Sequence Notes: †Related of | Subject<br>or unknown rela | AE reported | Preferre | d term | Grade | Relations | | Serious Event |
| Sequence Notes: † Related of Listing 10.1.2.3 | Subject<br>or unknown rela<br>3 Treatment di | AE reported ationship. | Preferre | d term | Grade<br>Adverse E | Relations) | | |
| Sequence Notes: † Related of Listing 10.1.2.3 | Subject or unknown rela 3 Treatment di Subject | AE reported ationship. Scontinuation d AE reported | Preferre<br>ue to non<br>Preferre | -related | Grade Adverse E Grade | Relationsl<br>vents<br>Relations | | |

Table 10.1.2.5 Reasons for study discontinuation

| S1 (TR) | | S2 (RT) | | Tota | 1 |
|---------|---|---------|---|------|---|
| N | % | N | % | N | % |

Patient's follow-up completed

Patient moved to Compassionate Use

Study termination

(clinical cut-off)

Withdrawal of consent

Death

Never treated

Lost to follow up

Other

Total

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### Listing 10.1.2.6 Reasons for study discontinuation due to other reason

| Sequence | Subject | Other, specify |
|---|---|---|
| Listing 10.1.2.7 Patients never treated | | |
| Sequence | Subject | Reason |

#### 10.1.3 Protocol Deviations

Classification will be based on the following group categories:

- Inclusion/exclusion criteria not met
- Incorrect treatment, dose or schedule received
- Excluded concomitant medication received
- Withdrawal criteria met, but treatment continued
- Failure to comply study procedures
- Any other Ethical/GCP issues

#### Listing 10.1.3.1 Relevant protocol deviations

| Sequence | Subject | Protocol deviation Type | Specify Deviation |
|----------|---------|-------------------------|-------------------|

#### 10.2 Patient Characteristics

Demographics and other baseline characteristics will be carried out on the enrolled population.

#### 10.2.1 Demographic and Other Baseline Characteristics

Table 10.2.1.1 Baseline characteristics: Gender

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

Gender

Male

Female

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.1.2 Baseline characteristics: Race

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

Race

White

Black

Asian

Other (Specify)

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.1.3 Baseline characteristics: Age

| | S1 (TR) | S2 (RT) | Total |
|----------------------|---------|---------|-------|
| Age at entry (years) | | | |

Ν

Mean, Std., Median, Range

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.1.4 Baseline characteristics: Pregnancy Test

| S1 (TR) | | S2 ( | RT) | Total | |
|---------|---|------|-----|-------|---|
| N | % | N | % | N | % |

Pregnancy Test

Positive

Negative

NA (Specify)

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

Table 10.2.1.5 Baseline characteristics: Adequate contraception

| S1 ( | TR) | S2 ( | RT) | То | tal |
|------|-----|------|-----|----|-----|
| N | % | N | % | N | % |

#### Adequate contraception

Yes

No

NA

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 10.2.2 Medical History

Listing 10.2.2.1 Ongoing medical history

| Sequence | Subject | Description | Onset date |
|----------|---------|-------------|------------|

#### 10.2.3 Cancer History

Table 10.2.3.1 First diagnosis: Tumor type

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

Tumor Type

Lung

Kidney

Prostate cancer

. . .

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.2 First diagnosis: Stage at diagnosis

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

Stage at Diagnosis

Early

Locally advanced

Metastatic

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

Table 10.2.3.3 First diagnosis: Time from first diagnosis to first infusion

S1 (TR) S2 (RT) Total Time form first diagnosis to first infusion (months) †

Mean, Std., Median, Range

Table 10.2.3.4 Current disease: Time from last PD to first infusion

| S1 (TR) | S2 (RT) | Total |
|---|---|---|
| Time from last PD <sup>†</sup> to first infusion (months) <sup>‡</sup> | | |

Mean, Std., Median, Range

Table 10.2.3.5 Current disease: Sites of disease involvement

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

Site of disease involvement

Lung

Liver

Lymph node

Pleura

Bone

Other (Specify)

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.6 No. of sites of disease involvement

| S1 ( | TR) | S2 (RT) | | Total | |
|------|-----|---------|---|-------|---|
| N | % | N | % | N | % |

No. of sites

1

2

 $\geq$  N sites

Total

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

<sup>†</sup> Time from first diagnosis to first infusion: defined as the date of first infusion minus date of first diagnosis.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Last PD will be taken from the Cancer history form

Firm from last PD to first infusion: defined as the date first infusion minus date of last progression before study

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.3.7 Summary statistics: No. of sites of disease involvement

| | S1 (TR) | S2 (RT) | Total |
|---|---|---|---|
| No. of sites | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test. | | | |

#### 10.2.4 Previous Anticancer Therapy Summary

Table 10.2.4.1 Patients with prior surgery

| S1 ( | TR) | S2 ( | RT) | То | tal |
|------|-----|------|-----|----|-----|
| N | % | N | % | N | % |

Prior surgery

Yes

No

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.2 Patients with prior radiotherapy

| S1 (TR) | | S2 ( | RT) | Total | |
|---------|---|------|-----|-------|---|
| N | % | N | % | N | % |

Prior radiotherapy

Yes

No

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.3 Prior anticancer medical therapy for study disease: No. of prior lines

| _ | S1 (TR) | | S2 (RT) | | Total | |
|---|---------|---|---------|---|-------|---|
| | N | % | N | % | N | % |

No. of prior lines

- 1 line
- 2 lines
- 3 lines
- >= 4 lines

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.4 Prior anticancer medical therapy for study disease: Summary of prior lines

| | S1 (TR) | S2 (RT) | Total |
|--------------------------------|---------|---------|-------|
| No. of prior lines | | | |
| N<br>Mean, Std., Median, Range | | | |

Table 10.2.4.5 Prior anticancer medical therapy for study disease: No. of prior chemotherapy lines

| 14010 10121110 11101 4111041001 111041041 1 | our merupy for study disease. It is of prior enemically miss | | | | | |
|---|---|---|---|---|---|---|
| | S1 (TR) | | S2 (RT) | | Total | |
| | N | % | N | % | N | % |
| No. of prior chemotherapy lines | | | | | | |
| 1 line | | | | | | |
| 2 lines | | | | | | |
| 3 lines | | | | | | |
| >= 4 lines | | | | | | |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.6 Prior anticancer medical therapy for study disease: Summary of prior chemotherapy lines

| Table 10.2.4.0 Filor anticancer medicar | merapy for study dise | ease. Summary of prio | i chemotherapy filles |
|---|---|---|---|
| | S1 (TR) | S2 (RT) | Total |
| No. of prior chemotherapy lines | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| S1, Sequence 1; S2, Sequence 2; TR, test-refe | erence; RT, reference-t | est. | |

Table 10.2.4.7 Prior anticancer medical therapy for study disease: No. of prior agents

| S1 (TR) | | S2 (RT) | | Total | |
|---------|---|---------|---|-------|---|
| N | % | N | % | N | % |

No. of prior agents

- 0 agents
- 1 agent
- 2 agents
- 3 agents

>= 4 agents

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.4.8 Prior anticancer medical therapy for study disease: Summary of prior agents

| | S1 (TR) | S2 (RT) | Total |
|---|---|---|---|
| No. of prior agents | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| S1. Sequence 1: S2. Sequence 2: TR. te | st-reference: RT. reference-te | st. | |

Table 10.2.4.9 Prior anticancer medical therapy for study disease: Time to progression of last therapy

| Time to progression (months) | S1 (TR) | S2 (TR) | Total |
|------------------------------|---------|---------|-------|
| N | | | |
| Mean, Std., Median, Range | | | |

### 10.2.5 Physical Examination, ECOG, Vital Signs, LVEF and ECG

| | Physical examination | | S1 (TR) | | S2 (RT) | | Total |
|---|---|---|---|---|---|---|---|
| Physical examir | action | N | % | N | % | N | % |
| Normal | | | | | | | |
| Abnormal | | | | | | | |
| | | er of patients in total<br>R, test-reference; RT, | | | applicable. | | |
| | | al examination: abr | normalities | | | | |
| Sequence | Subject | Description | | | | | |
| Γable 10.2.5.3 | Baseline physical | examination: Wei | ght, height a | and BSA | | | |
| Гable 10.2.5.3 | Baseline physical | examination: Wei | ght, height a | | 2 (RT) | Total | |
| Weight (kg) | Baseline physical | examination: Wei | | | 2 (RT) | Total | |
| Weight (kg)<br>N | | examination: Wei | | | 2 (RT) | Total | |
| Weight (kg)<br>N<br>Mean, Std., Me | | examination: Wei | | | 2 (RT) | Total | |
| Weight (kg)<br>N<br>Mean, Std., Me<br>Height (cm)<br>N | dian, Range | examination: Wei | | | 2 (RT) | Total | |
| Weight (kg)<br>N<br>Mean, Std., Me<br>Height (cm)<br>N<br>Mean, Std., Me | dian, Range | examination: Wei | | | 2 (RT) | Total | |
| Weight (kg)<br>N<br>Mean, Std., Me<br>Height (cm)<br>N<br>Mean, Std., Me<br>BSA (m <sup>2</sup> ) | dian, Range | examination: Wei | | | 2 (RT) | Total | |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me | dian, Range<br>dian, Range<br>dian, Range | | S1 (TR) | S: | 2 (RT) | Total | |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me | dian, Range<br>dian, Range<br>dian, Range | examination: Wei | S1 (TR) | S: | 2 (RT) | Total | |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me | dian, Range<br>dian, Range<br>dian, Range | | S1 (TR) | S: | 2 (RT) | Total | |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me S1, Sequence 1; | dian, Range dian, Range dian, Range S2, Sequence 2; TF | R, test-reference; RT, | S1 (TR) | S. | | Total | |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me SI, Sequence 1; | dian, Range dian, Range dian, Range S2, Sequence 2; TF | R, test-reference; RT, | S1 (TR) reference-tes | st. | s | | |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me S1, Sequence 1; | dian, Range dian, Range dian, Range S2, Sequence 2; TF | R, test-reference; RT, | S1 (TR) | st. | | | otal |
| Weight (kg) N Mean, Std., Me Height (cm) N Mean, Std., Me BSA (m²) N Mean, Std., Me S1, Sequence 1; | dian, Range dian, Range dian, Range S2, Sequence 2; TF | R, test-reference; RT, | S1 (TR) reference-tes | st. | s | | |

Notes: Percentage is based on number of patients in total and by sequence, when applicable. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

| Table | 10 2 5 5 | <b>Baseline</b> | characteristics: | Vital sions |
|--------|----------|-----------------|------------------|-------------|
| 1 auto | 10.2.3.3 | Dascillic | characteristics. | vitai signs |

| Table 10.2.3.3 Baseline characteris | | | |
|-------------------------------------|---------|---------|-------|
| | S1 (TR) | S2 (RT) | Total |
| Heart rate | | | |
| (Beats/minute) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| Temperature (°C) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| Blood pressure systolic (mmHg) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| Blood pressure diastolic | | | |
| (mmHg) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.5.6 Baseline characteristics: ECG<sup>†</sup> pre infusion

| | S1 (TR) | | S2 (RT) | | Total | | |
|-------------|---------|---|---------|---|-------|---|---|
| N % N % N % | N | % | N | % | | % | _ |

Result Normal Abnormal

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

† Worst result of the three ECGs replicates will be used as baseline value.

Table 10.2.5.7 Baseline characteristics: Pre infusion ECG<sup>†</sup> values

| | S1 | S1 (TR) | | S2 (RT) | | otal |
|---------------------------|----|---------|---|---------|---|------|
| | N | % | N | % | N | % |
| PR interval (msec) | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |
| Heart rate (bpm) | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |
| QT interval (msec) | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |
| Bazett's corrected QT | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |
| Fridericia's corrected QT | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |

<sup>†</sup> Mean of the three ECGs replicates will be used as baseline value.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.5.8 Baseline characteristics: Post-infusion ECG<sup>†</sup> values

| N | % | N | % | NI | 0./ |
|---|--------------|------------------------|-----------------------|----|-----|
| | | | 70 | N | % |
| | sed as hasel | sed as baseline value. | and an handling value | | |

Listing 10.2.5.9 Patients with abnormal electrocardiogram

| Sequence | Subject | ECG no. | Abnormality | PR interval (msec) | Heart rate (bpm) | QT interval (msec) | Bazett's corrected QT |
|---|---|---|---|---|---|---|---|
| , | | | | | | | |

Table 10.2.5.10 Baseline characteristics: LVEF

| S1 ( | TR) | S2 ( | RT) | То | otal |
|------|-----|------|-----|----|------|
| N | % | N | % | N | % |

Result

Normal

Abnormal

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 10.2.5.11 Patients with abnormal LVEF

| Sequence | Subject | Result | Method | Value (%) | Lower limit | Abnormalities |
|---|---|---|---|---|---|---|
| | | | | | (%) | |

Notes: Significant and non-significant abnormalities

Table 10.2.5.12 Baseline characteristics: LVEF value

| LVEF (%) by Method | S1 ( | (TR) | S2 ( | (RT) | Total | |
|---------------------------|------|------|------|------|-------|---|
| LVEF (%) by Method | N | % | N | % | N | % |
| MUGA | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |
| ЕСНО | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |
| Both | | | | | | |
| N | | | | | | |
| Mean, Std., Median, Range | | | | | | |

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

### 10.2.6 Hematological Evaluation at Baseline

Table 10.2.6.1 Hematology abnormalities at baseline<sup>†</sup>

| | | | S1 | (TR | .) | | | | S2 | (RT) | | | | | Tota | ıl | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | gr | All<br>ades | ( | Gr 1 | | •• | All g | rades | G | r 1 | | | gra | All<br>ides | G | r 1 | | |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| Anemia<br>Laukanania | | | | | | | | | | | | | | | | | | |

Leukopenia

Lymphopenia

Neutropenia

Thrombocytopenia

Table 10.2.6.2 Median and range for hematology parameters at baseline<sup>†</sup>

| Table 10.2.6.2 Median and range for | <u> </u> | | T 1 |
|---|---|---|---|
| | S1 (TR) | S2 (RT) | Total |
| Hemoglobin (g/dL) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| WBC (10%L) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| Lymphocytes (10%L) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| †Defined as the last value recorded before | e or on the date of first infusion | on. | |
| S1, Sequence 1; S2, Sequence 2; TR, test | -reference; RT, reference-tes | t. | |

Listing 10.2.6.3 Hematological abnormalities at baseline (grade  $\geq$  2)

| Sequence | Subject | Lab. Test | Examination date | Value | Unit | Std. Value | Std. Unit | Grade |
|---|---|---|---|---|---|---|---|---|

<sup>†</sup>Defined as the last value recorded before or on the date of first infusion.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

| Sequence | Subject | Lab. Test |
|----------|---------|-----------|
|----------|---------|-----------|

#### 10.2.7 Biochemical Evaluation at Baseline

Table 10.2.7.1 Biochemical abnormalities at baseline<sup>†</sup>

| | | S1 | (TR) | | | | S | S2 (R | (T) | | | | , | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | des | G | r 1 | | •• | | des | G | r 1 | | | | .ll<br>.des | Gı | r 1 | | |
| N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

ALT increased AST increased

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

| Table 10.2.7.2 Median and range for b | iochemical parameters a | t baseline <sup>†</sup> | |
|---|---|---|---|
| | S1 (TR) | S2 (RT) | Total |
| ALT (xULN) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| AST (xULN) | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| N | | | |
| Mean, Std., Median, Range | | | |
| †Defined as the last value recorded before | or on the date of first infusion | on. | |
| S1, Sequence 1; S2, Sequence 2; TR, test- | reference; RT, reference-tes | t. | |
| • | | | |
| Listing 10.2.7.2 Dischamical abnorma | liting at bagaling (anada) | > 2) | |

Listing 10.2.7.3 Biochemical abnormalities at baseline (grade  $\geq 2$ )

| Sequence | Subject | Lab. Test | Examination date | Value | Units | Std. Value | Std. Units | Grade | _ |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | _ |

#### Listing 10.2.7.4 Biochemical abnormalities not assessed at baseline

| Sequence | Subject | Lab. Test |
|----------|---------|-----------|

<sup>†</sup>Defined as the last value recorded before or on the date of first infusion.

<sup>\*</sup>Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia, hypocalcemia.

#### 10.2.8 Coagulation Evaluation at Baseline

Table 10.2.8.1 Coagulation abnormalities at baseline<sup>†</sup>

| | | S1 | (TR) | | | | S | S2 (R | .T) | | | | | Γotal | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| A<br>gra | | Gı | r 1 | | •• | | ll<br>des | Gı | r 1 | | | | ll<br>des | Gı | r 1 | | |
| <br>N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

INR increased

Listing 10.2.8.2 INR increased at baseline (grade  $\geq$  2)

| Sequence | Subject | Lab. Test | Examination date | Value | Std. Value | Grade |
|---|---|---|---|---|---|---|

#### Listing 10.2.8.3 INR not assessed at baseline

| Sequence | Subject | Lab. Test |
|----------|---------|-----------|

#### 10.2.9 Signs and Symptoms at Baseline

Signs and symptoms refer to any AE with onset date before the first treatment dose.

Table 10.2.9.1 Signs and symptoms at baseline (MedDRA coded)

| MedDRA SOC/PT <sup>†</sup> | S1 ( | TR) | S2 (1 | RT) | Total | |
|----------------------------|------|-----|-------|-----|-------|---|
| MCdDRA SOC/1 1 | N | % | N | % | N | % |
| | | | | | | • |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

Table 10.2.9.2 Signs and symptoms at baseline

| No. of signs and symptoms per | S1 (TR) | | S2 ( | (RT) | Total | |
|-------------------------------|---------|---|------|------|-------|---|
| patient | N | % | N | % | N | % |
| 0 | | | | | | |
| 1 | | | | | | |
| 2<br>≥ 3 | | | | | | |
| Total | | | | | | |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

Table 10.2.9.3 Summary of signs and symptoms at baseline

| No. of signs and symptoms per patient | S1 (TR) | S2 (RT) | Total |
|---------------------------------------|---------|---------|-------|

<sup>&</sup>lt;sup>†</sup>Defined as the last value recorded before or on the date of first infusion.

If INR increase is observed, check listing of concomitant medication (anticoagulants) in section 13

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup>SOC: System Organ Class; PT: Preferred Term

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

| No. of signs and symptoms per patient | S1 (TR) | S2 (RT) | Total |
|---|---|---|---|
| Mean, Std., Median, Range S1, Sequence 1; S2, Sequence 2; TR, test-refe | rence: RT reference-te | est | |
| 51, 564401100 1, 52, 564401100 2, 111, 1651 1610 | renee, ref, reference to | | |
| Listing 10.2.0.4 Ciana and assessed to | 1: (1- > 2) | | |

Listing 10.2.9.4 Signs and symptoms at baseline (grade  $\geq$  2)

| Sequence | Subject | Sign/symptom | MedDRA | Grade | Onset date | Relationship |
|---|---|---|---|---|---|---|
| | | | Preferred Term | | | |

#### 10.2.10 Concomitant Medication at Baseline

Concomitant medication at baseline according to the ATC classification.

Table 10.2.10.1 Concomitant medication at baseline (ATC levels1, 2 and 4)

| S1 (TR) | | S2 ( | RT) | Total | | |
|---------|---|------|-----|-------|---|---|
| N | % | N | % | N | % | _ |

Alimentary tract and metabolism
Antacids
Magnesium compounds
Magnesium adipate

. . .

Blood and blood forming organs Antithrombotic agents Vitamin K antagonists Acenocoumarol

. . .

Notes: Percentage is based on number of patients in total and by sequence, when applicable. S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 11 APPENDIX II: SAFETY ANALYSIS

Safety analysis will be carried out on evaluable patients for the safety population.

#### 11.1 Extent of exposure

#### 11.1.1 Treatment Administration

Table 11.1.1.1 Number of cycles administered<sup>†</sup>

| No. of a deciderate | S1 ( | S2 ( | S2 (RT) Total | | | |
|----------------------------|------|------|---------------|---|---|---|
| No. of cycles administered | N | % | N | % | N | % |
| 1 cycle | | | | | | |

<sup>2</sup> cycles

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

Table 11.1.1.2 Summary of number of cycles administered<sup>†</sup> and time on treatment

| Tuble 11:1:1:2 Building of Humber of ey | Tuble 11:1:12 Summary of number of cycles duministered and time on treatment | | |
|---|---|---|---|
| | S1 (TR) | S2 (RT) | Total |
| No. of cycles administered | | | |
| per patient | | | |
| N | | | |
| Median (range) | | | |
| Time on treatment (weeks)* | | | |
| N | | | |
| Median (range) | | | |

<sup>†</sup> Including when lurbinectedin is administered both alone and in combination with bosentan.

Table 11.1.1.3 Dose information by sequence

| | S1 (TR) | S2 (RT) | Total |
|-----------------------------|---------|---------------|-------|
| | | Lurbinectedin | |
| Cumulative dose (mg/m²) | | | |
| N | | | |
| Median (range) | | | |
| Dose intensity (mg/m²/week) | | · | |
| N | | | |
| Median (range) | | | |
| Relative dose intensity (%) | | | |
| N | | | |
| Median (range) | | | |
| | | Bosentan | |
| Cumulative dose (mg) | | | |
| N | | | |
| Median (range) | | | |

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>3</sup> cycles

<sup>†</sup> Including when lurbinectedin is administered both alone and in combination with bosentan.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>\*</sup>Time on treatment is defined as the last administration date of lurbinectedin plus 31 days, death or the start date of the new therapy, whichever comes first, minus the first administration date.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

### 11.1.2 Cycle Delays

Table 11.1.2.1 Summary of lurbinectedin dose delays

| | S1 ( | (TR) | S2 ( | (RT) | T | otal |
|---|---|---|---|---|---|---|
| _ | N | % | N | % | N | % |
| No. of patients treated | | | | | | |
| No. of patients susceptible to have dose delay | † | | | | | |
| No. of patients with any dose delay<br>Drug related <sup>‡</sup> AE<br>Non-drug related AE<br>Other reason | | | | | | |
| No. of cycles administered<br>No. of cycles susceptible to have dose delay <sup>††</sup> | | | | | | |
| No. of cycles with any dose delay <sup>‡</sup> Drug related <sup>‡</sup> AE Non-drug related AE Other reason | | | | | | |

<sup>†</sup> Excluding patients who received only the first cycle.

Table 11.1.2.2 Length of dosing delay

| S1 ( | TR) | S2 ( | RT) | Total | |
|------|-----|------|-----|-------|---|
| N | % | N | % | N | % |

#### Length of delay<sup>♯</sup>

Listing 11.1.2.3 Dose delays

| Sequence | Subject | Cycle | Delay (days) | Reason for delay |
|----------|---------|-------|--------------|------------------|

<sup>‡</sup> Related or unknown relationship

<sup>††</sup> All cycles excluding first cycle

<sup>†</sup> Denominator = Number of cycles susceptible to have dose delay S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

 $<sup>\</sup>leq$  7 days > 7 to  $\leq$  14 days

<sup>&</sup>gt; 14 days

Denominator = Number of cycles susceptible to have dose delay S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 11.1.3 Dose Reductions

Table 11.1.3.1 Summary of lurbinectedin dose reductions

| dosc rec | iuctions | | | | |
|---|---|---|---|---|---|
| S1 ( | (TR) | S2 ( | (RT) | То | otal |
| N | % | N | % | N | % |
| ion † | | | | | |
| n <sup>††</sup> | | | | | |
| 41 | | | | | |
| | S1 ( | S1 (TR) N % ion† | S1 (TR) S2 ( N % N ion† | S1 (TR) S2 (RT) N % N % ion† | N % N % N ion† |

<sup>†</sup> Excluding patients who received only the first cycle. ‡ Related or unknown relationship

Listing 11.1.3.2 Dose reductions

| Sequence | Subject | Cycle | Lurbinectedin intended dose (mg/m²) | Reason for dose reduction | Specify |
|---|---|---|---|---|---|

### 11.1.4 Any Other Dose Modifications

Listing 11 1 4 1 Dose interruptions for lurbinectedin

| Sequence Subject Cycl | | Cycle | Date | Reason for interruption | Specify |
|---|---|---|---|---|---|
| Listing 11.1.4. | 2 Dose not taken acco | ording to protoc | ol for Bose | ntan | |
| Sequence | Subject | | Cycle | Day | Reason |

<sup>††</sup> All cycles excluding first cycle

<sup>‡‡</sup> Denominator = Number of cycles susceptible to have dose delay/reduction

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 11.2 Adverse Events (AEs)

Adverse events tables will be listed by total and sequence or differentiating by treatment (Test, Reference or both).

Type of toxicity and worst grade or severity by cycle and by patient will be summarized according to System Organ Class (SOC) and Preferred Term (PT) as per the MedDRA dictionary. Subsequent grouping of similar or clinically related items might be appropriate at the time of the analysis.

Tables will be organized by category of events using SOC and PT. Grades could be presented by separate or any other grouping at the time of the analysis.

#### 11.2.1 Display of Adverse Events

Table 11.2.1.1 Summary of adverse events

| | LRB | LRB alone | |
|---|-----|-----------|---|
| N | % | N | % |

No. of patients with any AE

No. of patients with any treatment-related<sup>†</sup> AE

Patients with any grade  $\geq 3$  AE

Patients with any grade ≥4 AE

No. of patients with any grade  $\geq 3$  treatment-related<sup>†</sup> AE

No. of patients with any grade  $\geq 4$  treatment-related<sup>†</sup> AE

No. of patients with any SAE

No. of patients with any treatment-related † SAE

No. of patients with any grade  $\geq 3$  SAE

No. of patients with any grade ≥4 SAE

Any grade ≥3 treatment-related<sup>†</sup> SAE

Any grade ≥4 treatment-related<sup>†</sup> SAE

No. of patients with deaths associated with AEs

No. of patients with deaths associated with treatment-related<sup>†</sup> AEs

No. of patients with dose delays associated with AEs

No. of patients with dose delays associated with treatment-related<sup>†</sup> AEs

No. of patients with dose reductions associated with AEs

No. of patients with dose reductions associated with treatment-related<sup>†</sup> AEs

No. of patients with AEs leading to treatment discontinuation

No. of patients with treatment-related AEs leading to treatment discontinuation

Number of patients with at least one event, treatment modification, withdrawal or death during the treatment with BOS+LRB or LRB alone.

BOS, bosentan; LRB, lurbinectedin.

<sup>†</sup> Related to combination, lurbinectedin or bosentan, or with unknown relationship

Table 11.2.1.2 Treatment Related<sup>†</sup> (or with unknown relationship) Adverse Events. Worst grade per treatment

| | | BOS+LRB | | LRB alone | | |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | N % | N % | N % | N % | N % | N % |

. . .

Notes: Percentage is based on number of patients by treatment, when applicable.

† Related to both or lurbinectedin or bosentan or with unknown relationship

BOS, bosentan; LRB, lurbinectedin.

Table 11.2.1.3 Lurbinectedin related<sup>†</sup> Adverse Events. Worst grade per treatment

| | | BOS+LRB | | LRB alone | | |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | N % | N % | N % | N % | N % | N % |

..

Notes: Percentage is based on number of patients by treatment, when applicable.

† Related to lurbinectedin or with unknown relationship

BOS, bosentan; LRB, lurbinectedin.

Table 11.2.1.4 Bosentan related Adverse Events. Worst grade per treatment

| SOC/PT $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | | | BOS+LRB | |
|---|---|---|---|---|
| | SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | | N % | N % | N % |

..

Notes: Percentage is based on number of patients by treatment, when applicable.

† Related to bosentan or with unknown relationship

BOS, bosentan; LRB, lurbinectedin.

Table 11.2.1.5 Treatment Related<sup>†</sup> (or with unknown relationship) Adverse Events. Worst grade per

| patient | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S1 (TR) | | | | | S2 (RT) | | | | Total | | | | | | | |
| SOC/PT | | All<br>ides | Gr | ≥ 3 | Gr | ≥ 4 | | .ll<br>des | Gr | ≥3 | Gr | ≥4 | | des. | Gr | ≥ 3 | Gr | ≥4 |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

• • •

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

Table 11.2.1.6 Adverse Events regardless of relationship. Worst grade per treatment

| | BOS+LRB | | | LRB alone | | |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | Gr ≥ 4 | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | N % | N % | N % | N % | N % | N % |

..

Notes: Percentage is based on number of patients by treatment, when applicable.

BOS, bosentan; LRB, lurbinectedin.

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.
Table 11.2.1.7 Adverse Events regardless of relationship. Worst grade per patient

| | | | S1 | (TR) | | | | | S2 | (RT) | | | | | ] | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | | des. | Gr | ≥ 3 | Gr | ≥4 | All $Gr \ge 3$ $Gr \ge 4$ | | | | | ≥4 | All $Gr \ge 3$ $Gr \ge 4$ | | | | | ≥4 |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

# Listing 11.2.1.8 AEs grade $\geq 3$

| Sequence | Treatment | Cycle | Subject | SOC PT | Grade | SAE | Start | End | Relationship | Action | Serious | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group <sup>†</sup> | | | | | (Y/N) | date | date | study | taken | Event | |
| | | | | | | | | | medication | | | |

## †BOS+LRB/LRB alone

#### Listing 11.2.1.9 AEs related only to lurbinectedin

| Sequence | Treatment | Cycle | Subject | SOC | PT | Grade | SAE | Start | End | Action | Serious | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | group <sup>†</sup> | | | | | | (Y/N) | date | date | taken | Event | |

<sup>†</sup>BOS+LRB/LRB alone

#### Listing 11.2.1.10 AEs related only to bosentan

| Sequence | Treatment | Cycle | Subject | SOC | PT Grade | SAE | Start | End | Action | Serious | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | group <sup>†</sup> | | | | | (Y/N) | date | date | taken | Event | |

<sup>†</sup>BOS+LRB

#### 11.3 Serious Adverse Events and Deaths

#### 11.3.1 Serious Adverse Events

Serious adverse events tables will be listed by total and sequence or differentiating by treatment (Test, Reference or both).

Type of toxicity and worst grade or severity by cycle and by patient will be summarized according to System Organ Class (SOC) and Preferred Term (PT) as per the MedDRA dictionary. Subsequent grouping of similar or clinically related items might be appropriate at the time of the analysis.

Tables will be organized by category of events using SOC and PT. Grades could be presented by separate or any other grouping at the time of the analysis.

If the number of SAEs are very low, these tables will not be presented and only listings will be shown.

Table 11.3.1.1 Treatment Related† (or with unknown relationship) SAEs. Worst grade per treatment

| | | BOS+LRB | | L | RB alone | |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | N % | N % | N % | N % | N % | N % |

Notes: Percentage is based on number of patients by treatment, when applicable.

BOS, bosentan; LRB, lurbinectedin.

Table 11.3.1.2 Lurbinectedin related<sup>†</sup> SAEs. Worst grade per treatment

| | | BOS+LRB | | L | RB alone | |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| SOC/P1 | N % | N % | N % | N % | N % | N % |

Notes: Percentage is based on number of patients by treatment, when applicable.

BOS, bosentan; LRB, lurbinectedin.

Table 11.3.1.3 Bosentan related<sup>†</sup> SAEs. Worst grade per treatment

| | | | BOS+LRB | | | |
|--------|---------|-----|---------|-----|----|----|
| SOC/DT | All gra | des | Gr 2 | ≥ 3 | Gr | ≥4 |
| SOC/P1 | N | % | N | % | N | % |

Notes: Percentage is based on number of patients by treatment, when applicable.

BOS, bosentan; LRB, lurbinectedin.

Table 11.3.1.4 Treatment Related† (or with unknown relationship) SAEs. Worst grade per patient

| | | S1 (TR) | | | | | | | S2 | | ) | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | All<br>grades Gr≥ | | ≥3 | $Gr \ge 4$ | | All<br>grades | | Gr | ≥ 3 | $Gr \ge 4$ | | | des | Gr | ≥ 3 | Gr | ≥4 | |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship

<sup>†</sup> Related to lurbinectedin or with unknown relationship

<sup>†</sup> Related to bosentan or with unknown relationship

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.3.1.5 SAEs regardless of relationship. Worst grade per treatment

| | | BOS+LRB | | | LRB | alone |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| | N % | N % | N % | N % | N % | N % |

. . .

Notes: Percentage is based on number of patients by treatment, when applicable. BOS, bosentan; LRB, lurbinectedin..

Table 11.3.1.6 SAEs regardless of relationship. Worst grade per patient

| | | S1 (TR) | | | | | | S2 | (RT | ) | | | | Total | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | A<br>grad | | Gr | ≥ 3 | Gr | ≥4 | A<br>gra | ll<br>des | Gr | ≥ 3 | Gr | ≥4 | | ll<br>des | Gr | ≥3 | Gr | ≥4 |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

. . .

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.3.1.7 All SAEs<sup>†</sup>

| Sequence Treatment Cycle | Subject | SOC PT | Grade | ΑE | AE | AE | Start | End date |
|---|---|---|---|---|---|---|---|---|
| group* | | | | Status | Relationship | consequences | date | |

<sup>†</sup> SAE narratives will be provided by the pharmacovigilance department

#### 11.3.2 Deaths

Table 11.3.2.1 Cause of death

| S1 ( | TR) | 82.6 | RT) | Total | |
|------|-----|------|-----|-------|---|
| N | % | N | % | N | % |

Malignant disease

Adverse Event(s)

Other<sup>‡</sup>

Total

Notes: Percentage is based on number of patients who died by total and sequence, when applicable.

Listing 11.3.2.2 Deaths

| Listing 11.5. | 2.2 Deaths | | | | | |
|---|---|---|---|---|---|---|
| Sequence | Subject | Death date | Cause of | No. of cycles | Time on treatment <sup>†</sup> | Time from last |
| | | | death | administered | | dose‡ (days) |

<sup>†</sup> Time on treatment is defined as the last administration date of lurbinectedin plus 31 days, death or the start date of the new therapy, whichever comes first, minus the first administration date.

<sup>\*</sup>BOS+LRB/LRB alone

<sup>‡</sup> Specify

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>&</sup>lt;sup>‡</sup>Time from last dose defined as date of death minus date of last infusion.

# 11.4 Clinical Laboratory Evaluation

# 11.4.1 Hematological Abnormalities

| | | BOS | +LRB | | | | | | LRB a | lone | ; |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | All grade | s Gr | ≥ 3 | Gr≥4 | | All g | grades | G | $r \ge 3$ | Gr | ≥4 |
| | N % | N | % | N % | | N | % | N | I % | N | % |
| nemia | | | | | | | | | | | |
| eukopenia | | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | | |
| Veutropenia | | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | | |
| lotes: Percentage is bas | ad an numbar | of notiont | a hritman | tmant rich | on annlica | hla | | | | | |
| | | or patient | s by nea | imeni, wii | еп аррпса | bie. | | | | | |
| BOS, bosentan; LRB, lu | ii dinectedin. | | | | | | | | | | |
| Listing 11.4.1.2 Hema | | normaliti | es grad | | | | | | | | |
| Treatment | Subject | | | Event | | | Gra | de | | | |
| group <sup>†</sup> | | | | | | | | | | | |
| BOS+LRB/LRB alone | | | | | | | | | | | |
| POD - PICD/ PICD GIVIIC | | | | | | | | | | | |
| Listing 11.4.1.3 Hema | atological test | ts not ass | sessed b | y patient | | | | | | | |
| Treatment | | Subject | | | | Lab. t | est | | | | |
| group <sup>†</sup> | | 3 | | | | | | | | | |
| BOS+LRB/LRB alone | | | | | | | | | | | |
| | ological abno | ormalitie | s: Wors | t grade pe | er patient | | | | | | |
| | ological abno | ormalitie:<br>S1 (TR) | | | er patient<br>S2 (RT) | | | | Total | | |
| | ological abno | S1 (TR) | | | S2 (RT) | | A | | | | |
| | | | | | _ | Gr ≥ 4 | A<br>gra | | $Total$ $Gr \ge 3$ | G | ìr≥ |
| | All | S1 (TR) | | All<br>grades | S2 (RT) | | gra | | | G | |
| <u>Γable 11.4.1.4 Hemat</u> | All grades | S1 (TR) $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $\frac{\text{S2 (RT)}}{\text{Gr} \ge 3}$ | Gr ≥ 4 | gra | des | Gr ≥ 3 | | |
| Γable 11.4.1.4 Hemat | All grades | S1 (TR) $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $\frac{\text{S2 (RT)}}{\text{Gr} \ge 3}$ | Gr ≥ 4 | gra | des | Gr ≥ 3 | | |
| Γable 11.4.1.4 Hemat Anemia Leukopenia | All grades | S1 (TR) $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $\frac{\text{S2 (RT)}}{\text{Gr} \ge 3}$ | Gr ≥ 4 | gra | des | Gr ≥ 3 | | |
| Table 11.4.1.4 Hemat Anemia Leukopenia Lymphopenia | All grades | S1 (TR) $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $\frac{\text{S2 (RT)}}{\text{Gr} \ge 3}$ | Gr ≥ 4 | gra | des | Gr ≥ 3 | | |
| Anemia Leukopenia Lymphopenia Neutropenia | All grades | S1 (TR) $Gr \ge 3$ | Gr ≥ 4 | All<br>grades | $\frac{\text{S2 (RT)}}{\text{Gr} \ge 3}$ | Gr ≥ 4 | gra | des | Gr ≥ 3 | | |
| Table 11.4.1.4 Hemat Anemia Leukopenia Lymphopenia Neutropenia Chrombocytopenia | All<br>grades<br>N % | S1 (TR) Gr ≥ 3 N % | Gr ≥ 4<br>N % | All grades | S2 (RT) Gr ≥ 3 N % | Gr ≥ 4<br>N % | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Fable 11.4.1.4 Hemat Anemia Leukopenia Lymphopenia Neutropenia Notes: Percentage is bas | All grades N % | $S1 (TR)$ $Gr \ge 3$ $N$ % | $Gr \ge 4$ $N = \%$ s in total | All grades N % | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, w | Gr ≥ 4<br>N % | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Anemia Leukopenia Lymphopenia Neutropenia Thrombocytopenia Notes: Percentage is bas | All grades N % | $S1 (TR)$ $Gr \ge 3$ $N$ % | $Gr \ge 4$ $N = \%$ s in total | All grades N % | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, w | Gr ≥ 4<br>N % | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Anemia Leukopenia Lymphopenia Neutropenia Thrombocytopenia Notes: Percentage is bas | All grades N % | $S1 (TR)$ $Gr \ge 3$ $N$ % | $Gr \ge 4$ $N = \%$ s in total | All grades N % | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, w | Gr ≥ 4<br>N % | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Table 11.4.1.4 Hemat Anemia Leukopenia Lymphopenia Neutropenia Γhrombocytopenia | All grades N % | $S1 (TR)$ $Gr \ge 3$ $N$ % | $Gr \ge 4$ $N = \%$ s in total | All grades N % | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, w | Gr ≥ 4<br>N % | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Anemia Leukopenia Lymphopenia Neutropenia Fhrombocytopenia Notes: Percentage is bas S1, Sequence 1; S2, Seq | All grades N % | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ s in tota nce; RT, | All grades N % and by se | $S2 (RT)$ $Gr \ge 3$ $N \%$ equence, we-test. | Gr ≥ 4<br>N % | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Anemia Leukopenia Lymphopenia Neutropenia Notes: Percentage is bas S1, Sequence 1; S2, Sequenc | All grades N % sed on number quence 2; TR, to | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ As in total ance; RT, | All grades N % and by se reference- | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |
| Anemia Leukopenia Lymphopenia Neutropenia Notes: Percentage is bas S1, Sequence 1; S2, Sequenc | All grades N % | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ s in tota nce; RT, | All grades N % and by se reference- | $S2 (RT)$ $Gr \ge 3$ $N \%$ equence, we-test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3 | | |
| Anemia Leukopenia Lymphopenia Neutropenia Notes: Percentage is bas S1, Sequence 1; S2, Sequenc | All grades N % sed on number quence 2; TR, to | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ As in total ance; RT, | All grades N % and by se reference- | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |
| Anemia Leukopenia Lymphopenia Neutropenia Notes: Percentage is bas S1, Sequence 1; S2, Sequenc | All grades N % sed on number quence 2; TR, to | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ As in total ance; RT, | All grades N % and by se reference- | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |
| Anemia Leukopenia Lymphopenia Neutropenia Notes: Percentage is bas S1, Sequence 1; S2, Sequenc | All grades N % sed on number quence 2; TR, to | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ As in total ance; RT, | All grades N % and by se reference- | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |
| Anemia Leukopenia Lymphopenia Leutropenia Lotes: Percentage is bas L1, Sequence 1; S2, Sequenc | All grades N % sed on number quence 2; TR, to | $S1 (TR)$ $Gr \ge 3$ $N \%$ of patient est-reference | $Gr \ge 4$ $N = \%$ As in total ance; RT, | All grades N % and by se reference- | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |
| nemia eukopenia ymphopenia leutropenia hrombocytopenia lotes: Percentage is bas 1, Sequence 1; S2, Seq isting 11.4.1.5 Hema equence Si | All grades N % sed on number quence 2; TR, to atological abrubject | $S1 (TR)$ $Gr \ge 3$ $N$ % of patient est-reference to the company of the company | $Gr \ge 4$ $N = \%$ s in tota nce; RT, es by cy Eve | All grades N % and by se reference- vele gradent | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |
| Anemia Leukopenia Lymphopenia Notes: Percentage is bas S1, Sequence 1; S2, Seq Listing 11.4.1.5 Hema Sequence Listing 11.4.1.6 Hema | All grades N % sed on number quence 2; TR, to atological abrubject | $S1 (TR)$ $Gr \ge 3$ $N$ % of patient est-reference to the companion of th | Gr ≥ 4 N % s in tota nce; RT, es by cy Eve | All grades N % and by se reference- vele gradent | $\begin{array}{c} \text{S2 (RT)} \\ \text{Gr} \geq 3 \\ \text{N} \% \\ \\ \text{equence, w-test.} \\ \\ \text{e} \geq 3 \\ \text{Cycle} \end{array}$ | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | Gr ≥ . |
| Anemia Leukopenia Lymphopenia Notes: Percentage is bas S1, Sequence 1; S2, Seq Listing 11.4.1.5 Hema Sequence Listing 11.4.1.6 Hema | All grades N % sed on number quence 2; TR, to atological abrubject | $S1 (TR)$ $Gr \ge 3$ $N$ % of patient est-reference to the company of the company | Gr ≥ 4 N % s in tota nce; RT, es by cy Eve | All grades N % and by se reference- vele gradent | $S2 (RT)$ $Gr \ge 3$ $N %$ equence, we test. | $Gr \ge 4$ $N = \frac{9}{2}$ Then app | gra<br>N | des<br>% | Gr ≥ 3<br>N % | | |

#### 11.4.2 Biochemical Abnormalities

| All grades $Gr \ge 3$ $Gr \ge 4$ All grades $Gr \ge 3$ $Gr \ge 4$ | | BOS+LRE | 3 | LRB alo | | |
|---|---|---|---|---|---|---|
| N 0/ N 0/ N 0/ N 0/ N 0/ N 0/ N 0/ | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| N % N % N % N % N % N % | N % | N % | N % | N % | N % | N % |

ALT increase AST increase

. . . . 4

Notes: Percentage is based on number of patients by treatment, when applicable.

\*Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypercalcemia, hypocalcemia.

BOS, bosentan; LRB, lurbinectedin.

Listing 11.4.2.2 Biochemical abnormalities grade  $\geq 3$ 

| | | <i>0</i> ···· <u> </u> | |
|--------------------|---------|------------------------|-------|
| Treatment | Subject | Event | Grade |
| group <sup>†</sup> | | | |

†BOS+LRB/LRB alone

Listing 11.4.2.3 Biochemical tests not assessed

| Treatment | Subject | Lab. test |
|--------------------|---------|-----------|
| group <sup>†</sup> | • | |

†BOS+LRB/LRB alone

Table 11.4.2.4 Biochemical abnormalities: Worst grade per patient

| S1 (TR) | | | | | S2 (RT) | | | | | Total | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| All grades Gr≥3 C | | Gr | ≥4 | $ \begin{array}{cc} \text{All} & \text{Gr} \ge 3 \\ \text{grades} & \text{Gr} \ge 3 \end{array} $ | | ≥ 3 | $Gr \ge 4$ All grades | | | | Gr | ≥ 3 | Gr | ≥4 | | | |
| N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

ALT increase AST increase

...\*

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

\*Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypercalcemia, hypocalcemia

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Listing 11.4.2.5 Biochemical abnormalities by cycle grade  $\geq 3$ 

| Sequence | Subject | Event | Cycle | Grade |
|----------|---------|-------|-------|-------|

Listing 11.4.2.6 Biochemical tests not assessed by cycle

| Sequence | Subject | Cycle | Lab. test |
|----------|---------|-------|-----------|

# 11.4.3 Laboratory Values Over Treatment

Table 11.4.3.1 Shift of hematological abnormalities, worst grade per patient vs. baseline

| | - | | | Wors | st grade | per pat | ient dur | ing trea | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | Gra | de 1 | | de 2 | | de 3 | | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | S1 | (TR) | | | | |
| Anemia | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| Leukopenia | Grade 0 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| * | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| | | | | | | S2 | (RT) | | | | |
| Anemia | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| Leukopenia | Grade 0 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| * | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| | | | | | | To | otal | | | | |
| Anemia | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| Leukopenia | Grade 0 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| * | Grade 0 | | | | | | | | | | |
| | ••• | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

If a low number of patients with grade  $\geq 3$  neutropenia or thrombocytopenia, the following table will be omitted and the information will be provided in a listing.

Table 11.4.3.2 Time course for neutrophils and platelets

| | В | BOS+LRB | | 3 alone | | Total |
|---|---|---|---|---|---|---|
| | N | Median<br>(range) | N | Median<br>(range) | N | Median (range) |
| Neutropenia (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Nadir day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |
| Thrombocytopenia (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Nadir day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |

<sup>\*</sup>Lymphopenia, Neutropenia and Thrombocytopenia.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.4.3.3 Shift of biochemical abnormalities, worst grade per patient vs baseline

| | int of blochemical abi | | | | | | tient du | | tment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline grade | Gra | | Gra | de 2 | Gra | ide 3 | Gra | de 4 | Gra | de 5 |
| | | N | % | N | % | N | % | N | % | N | % |
| | | | | | | S1 | (TR) | | | | |
| ALT increase | Grade 0 | | | | | | | | | | |
| . am : | Grade 4 | | | | | | | | | | |
| AST increase | Grade 0 | | | | | | | | | | |
| at. | Grade 4 | | | | | | | | | | |
| * | Grade 0 | | | | | | | | | | |
| | <br>C 1- 4 | | | | | | | | | | |
| | Grade 4 | | | | | G2 | (DT) | | | | |
| | | | | | | S2 | (RT) | | | | |
| ALT increase | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| AST increase | Grade 0 | | | | | | | | | | |
| ala. | Grade 4 | | | | | | | | | | |
| * | Grade 0 | | | | | | | | | | |
| | <br>Cm. d. 4 | | | | | | | | | | |
| | Grade 4 | | | | | T | . 1 | | | | |
| | | | | | | 10 | otal | | | | |
| ALT increase | Grade 0 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |
| AST increase | Grade 0 | | | | | | | | | | |
| ala. | Grade 4 | | | | | | | | | | |
| * | Grade 0 | | | | | | | | | | |
| | <br>Cando 4 | | | | | | | | | | |
| | Grade 4 | | | | | | | | | | |

Notes: Percentage is based on number of patients in total and by sequence, when applicable.

If a low number of patients with grade  $\geq 3$  ALT or AST increased, the following table will be omitted and the information will be provided in a listing.

Table 11.4.3.4 Time course for AST and ALT

| | В | OS+LRB | LR | B alone | Total | |
|---|---|---|---|---|---|---|
| | N | Median<br>(range) | N | Median<br>(range) | N | Median<br>(range) |
| AST (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Peak day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |
| ALT (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Peak day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |
| BOS bosenton: I DR Jurbinectedin | | | | | | |

<sup>†</sup>For ALT, AST, AP, GGT, and Bilirubin parameters, worst grade will be calculated compared to baseline.

<sup>\*</sup>Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased,

hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypocalcemia, hypocalcemia.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

If appropriate, inter-cycle time courses for neutropenia, thrombocytopenia or any other significant parameter will be displayed in graphs.

## 11.5 Linear Mixed-effects Model

If applicable, to compare the incidence of grade  $\geq 4$  or grade  $\geq 3$  between the combination and lurbinectedin alone, a generalized linear mixed-effects model will be fit to the data with treatment (Combination or lurbinectedin alone), period and sequence as fixed effects, and patients nested in sequences as a random effect.

Table 11.5.1.1 Safety comparison between combination and lurbinectedin alone<sup>†</sup>

| | Combination | Lurbinectedin alone | p-value‡ |
|---|---|---|---|
| Any grade ≥3AE | | | |
| Any grade ≥4 AE | | | |
| Any grade ≥3 treatment-related AE | | | |
| Any grade ≥4 treatment-related AE | | | |
| Any abnormality $(G \ge 3)$ in | | | |
| laboratory value (hema, bio) | | | |
| Any abnormality (G≥4) in | | | |
| laboratory value (hema_bio) | | | |

<sup>†</sup> A generalized mixed-effects model will be fit for each safety evaluation

# 11.6 Physical Findings, ECOG PS, LVEF and ECG

#### 11.6.1 Physical Findings and ECOG PS

Listing 11.6.1.1 ECOG Performance status during the study

| Sequence | Subject | | | $\mathrm{PS}^{\dagger}$ | | |
|---|---|---|---|---|---|---|
| | 3 | Baseline | Cycle 1 | Cycle 2 | Cycle 3 | EOT |
| S1 (TR) | ••• | | | | | |
| S2 (RT) | | | | | | |

<sup>†</sup> Worst of cycle determination

Listing 11.6.1.2 Weight change during the study

| | | | | % Change <sup>†</sup> | | |
|---|---|---|---|---|---|---|
| Sequence | Subject | Weight at<br>Baseline | Cycle 1 | Cycle 2 | Cycle 3 | EOT |
| S1 (TR) | | | | | | |
| S2 (RT) | | | | | | |

<sup>†%</sup> compared to baseline

#### 11.6.2 LVEF and ECG

Listing 11.6.2.1 Patients with abnormal or clinically indicated LVEF during the study

| 0 | | | | | 0 | | |
|---|---|---|---|---|---|---|---|
| Sequence | Subject | Assessment Date | Abnormality | Specify | Method | LVEF | Lower limit of |
| | | | | | | (%) | normality |

<sup>‡</sup>p-values will be provided for the comparison between treatments (combination vs. Lurbinectedin alone) or including the sequence effect if deemed necessary.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

| Sequence | Subject | Assessment Date | Abnormality | Specify | Method | LVEF<br>(%) | Lower limit of normality |
|---|---|---|---|---|---|---|---|

Listing 11.6.2.2 Electrocardiogram evolution during the study

| Sequence | Subject | % Change <sup>†</sup> | | | | | |
|---|---|---|---|---|---|---|---|
| | _ | ECG<br>parameters*<br>Baseline | Cycle 1<br>Pre infusion | Cycle 1<br>Post infusion | Cycle 2<br>Pre infusion | Cycle 2<br>Post infusion | ЕОТ |
| S1 (TR) | ••• | | | | | | |
| S2 (RT) | | | | | | | |

<sup>\*</sup> PR interval (msec), Heart rate (bpm), QT interval (msec), QRS complex duration, Fridericia corrected QT  $^{\dagger}$ % compared to baseline

Listing 11.6.2.3 Patients with abnormal or clinically indicated Electrocardiogram during the study

| | | | | | | | | <u> </u> |
|---|---|---|---|---|---|---|---|---|
| Sequence | Subject | Assessment Date | Result | Specify | PR | Heart | QT | Bazett's |
| | | | | | Interval | rate (bpm) | interval | corrected QT |
| | | | | | (msec) | | (msec) | |

# 11.7 Concomitant Therapies

## 11.7.1 Concomitant Medication during the Study

Table 11.7.1.1 Concomitant medication during treatment (ATC1/ATC2/ATC4/PN)

| | BOS+LRB | LRB alone |
|---------------------------------|---------|-----------|
| | N % | N % |
| Alimentary tract and metabolism | | |
| Antacids | | |
| Magnesium compounds | | |
| Magnesium adipate | | |
| Blood and blood forming organs | | |
| Antithrombotic agents | | |
| Vitamin K antagonists | | |
| Acenocoumarol | | |

Notes: Percentage is based on number of patients by treatment, when applicable. BOS, bosentan; LRB, lurbinectedin.

<sup>&</sup>lt;sup>‡</sup> Triplicate ECG values obtained at each time point (baseline, Day 1 of Cycle 1 pre-infusion and post-infusion, Day 1 of Cycle 2 pre-infusion and post-infusion and end of treatment) are averaged

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.7.1.2 Summary of concomitant medication during treatment by ATC

| Table 11.7.1.2 Summary of concomitant medication | | | | |
|---|---|---|---|---|
| | BOS+ | -LRB | LRB a | llone |
| | N | % | N | % |
| No. of systems (ATC1 level) | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| ≥ 3 | | | | |
| Median (range) | | | | |
| No. of indications (ATC2 level) | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| $\geq 3$ | | | | |
| Median (range) | | | | |
| No. of agent families (ATC4 level) | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| ≥3 | | | | |
| Median (range) | | | | |
| No. of agents (PN level) | | | | |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| ≥ 3 | | | | |
| Median (range) | | | | |

# BOS, bosentan; LRB, lurbinectedin.

# 11.7.2 Further Antitumor Therapies

Listing 11.7.2.1 First Antitumor Therapy

| Sequence | ence Subject End of treatment | First Antitumor Therapy | Start date |
|---|---|---|---|

# 12 APPENDIX III: EFFICACY ANALYSIS

Not applicable.

# 13 APPENDIX IV: DB Listings

| Listing 13. | 1 Screenii | ng (I) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Sequence | Subject | Informed consent | PGt<br>sub-study | Planned initiation | | EC4 | PCR date | PCR result | Eligibility |
| Listing 13. | 2 Screenii | ng (II) | | | | | | | |
| Sequence | 2 201001111 | Subject | | Screening f | ailure | | Criteri | on not met | Details |
| Listing 13. | 3 Study re | egistration/Ra | andomizati | on details | | | | | |
| Sequence | Subject | Rando | mization D | | | Treatm | | eatment | Screening |
| | | | K | andomizatio | 11 , | Sequen | ce De | scription | failure date |
| Listing 13. | 4 Date of | visit | | | | | | | |
| Se | equence | | Subject | | | Visi | it | | Date |
| | | unscheduled | | *** | | | | | 11 1 11 1 |
| Sequ | ence | Subje | ect | Visit | i | | Date | Clini | cally indicated repeat |
| | | | | | | | | | Topeat |
| Listing 13. | | | | | | | | | |
| Sequence | Subje | ct Dat | te of birth | Age Deriv (years) | ed | Sex | Race | Other Ra | ce, specify |
| | | | | (years) | | | | | |
| Listing 13. | 7 Childbe | aring potenti | | _ | aceptio | n | | | |
| Sequence | Subject | Childb | earing pote | | - | A | dequate cont | raception? | Specify |
| | | | | Rea | SOII | | | | |
| Listing 13. | 8 Pregnan | icy test | | | | | | | |
| Sequence | Subject | | pplicable? | Reas | son | Not do | one? | Sample date | Result |
| | | edical history | | OC M | ADDA | DT | On set data | Resolve | d On a sin a |
| Sequence | Subject | Descripti | ion S | OC Me | edDRA : | PI | Onset date | date | d Ongoing |
| | 10.0 | • • • | | | | | | | |
| Listing 13. | 10 Cancer | r history | First dia | anogia | | | Current | diganga | |
| Sequence | Subject | Date of | Tumor | | te of | | Date of | | te of Sites |
| Sequence | Buoject | diagnosis | type | U | vanced o | disease | | | PD |
| | | | | | | | | | <u> </u> |
| Listing 12 | 11 Drior a | urgary | | | | | | | |
| Listing 13. Sequence | 11 PHOI S | Subject | N | one? | | Site | and procedur | res | Date |
| zequence | | 240,000 | 1 | | | 5110 | a procedu | | _ *** |
| | | adiotherapy | C: | | 1.1. | (C.) | D : 07 | . 1 = | |
| Sequence | Subject | None? | Site<br>(Anato | | ıl dose ( | Gy) | Date of firs | t dose Da | te of last dose |
| | | | (Anatt | 11110) | | | | | |

| Sequence | Subject | None? | Regimen | Agent | Agent<br>Coded | Agent<br>Class | Setting | Start S<br>date o | _ | Best<br>response | | Non PD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | hylactic m | | | | | | | | | | |
| Sequence | Subject | Visit Typ | e Medicat | ion† | | Daily Ui<br>lose | | Start Sto<br>late dat | _ | me Take<br>prote | _ | Specify |
| (†) ATC1, | ATC2, AT | C3, ATC4 | | | | | | | | | | |
| | | inectedin a | | ation | | | | | | | | |
| Sequence | Subject V | isit Date | Route | Start<br>time | time d | ntended<br>lose<br>mg/m²) | Total i<br>dose (1 | | Fotal<br>lose<br>given | Total<br>volume | | A<br>culated<br>dose |
| Listing 1 | 3.16 Lurb | inectedin t | reatment | modifi | cation | | | | | | | |
| Sequence | Subject | Visit | Any mo | | on Treat | ment | Reas | son Ac | dverse | Event ( | Other, s | specify |
| | | | | | WIOU | incation | | | | | | |
| Listing 1. | 3.17 Lurb | inectedin r | e-admini | stration | 1 | | | | | | | |
| Sequence | Subject | Visit | Date | e l | Not done? | Rout | e Tota | ıl dose gi | ven S | Start time | End | time |
| | | ntan admii | | | | | | | | | | |
| | | ntan admii<br>Visit Day | | prior t<br>Time | | capsules | Taken | I<br>lingly? | Reasor | n Conta | No | 0 |
| Sequence | Subject | Visit Day | Date | Time | No. of 6<br>(125 m) | capsules | Taken | | Reasor | n Conta | No | 0 |
| Sequence Listing 1. | Subject 3.19 Hem | Visit Day | Date | Time y value | No. of o<br>(125 m | capsules | Taken<br>accord | lingly? | | n Conta | No<br>co | 0 |
| Sequence Listing 1: Sequence | Subject 3.19 Hem Subject | Visit Day atological Calc. Da | laborator | Time y value | No. of o<br>(125 m | capsules<br>g) | Taken<br>accord | lingly? | s Lyr | | No co | o<br>ntacted |
| Sequence Listing 1: Sequence | Subject 3.19 Hem Subject | Visit Day<br>atological<br>Calc. Da | laborator | Time y value | No. of o<br>(125 m | capsules<br>g)<br>WB | Taken<br>accord | lingly? | s Lyr | nphocyte | No co | ontacted |
| Sequence Listing 1: Sequence (†) Hemato | Subject 3.19 Hem Subject Decrit, RBC | Visit Day atological Calc. Da | laborator<br>ite Hem<br>(§ | Time y value | No. of 6 (125 mg | wB | Taken<br>accord | lingly? | s Lyr | nphocyte | No co | ontacted |
| Listing 1: Sequence (†) Hemato | 3.19 Hem Subject Decrit, RBC | atological Calc. Day | laborator<br>ite Hem<br>(§ | Time y value oglobin y/dl) | No. of o<br>(125 m | wB | Taken<br>accord | lingly?<br>eutrophil<br>x10*9/L) | s Lyr | mphocyte<br>(10*9/L) | No co | telets<br>0*9/L) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence | 3.19 Hem<br>Subject<br>Derit, RBC<br>3.20 Coag | atological Calc. Da cycle and monoc gulation Te | laborator tte Hem (g ytes. | Time<br>y value<br>oglobin<br>g/dl) | No. of c<br>(125 mg | wB | Taken<br>accord<br>BC N<br>9/L) ( | lingly?<br>eutrophil<br>x10*9/L) | s Lyı | mphocyte<br>(10*9/L) | s Pla (x10 | o<br>ntacted<br>telets<br>)*9/L) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence | 3.19 Hem<br>Subject<br>Derit, RBC<br>3.20 Coag | atological Calc. Da cycle and monocy gulation Te Subject hemical lal isit Calc. | laborator tte Hem (g ytes. | Time y value oglobin y/dl) values Total | No. of c (125 m) es† Calculate cycle | wB (x10* | Taken accord | eutrophil<br>x10*9/L) | s Lyr<br>(x<br>epeat | nphocyte<br>(10*9/L) | s Pla (x10 | telets<br>0*9/L) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence Listing 1: Sequence | 3.19 Hem Subject Subject Subject 3.20 Coag 3.21 Bioci | atological Calc. Da cycle and monocy gulation Te Subject hemical la isit Calc. Cycle | laborator tte Hem (g ytes. St Visit boratory Date n | Time y value oglobin g/dl) values Total (mg/ | No. of c (125 m) es† Calculate cycle I Bilirubin dl) | wB (x10* | Taken accord | eutrophil<br>x10*9/L) | s Lyr<br>(x<br>epeat | nphocyte (10*9/L) I LT LI U/L) (x | s Pla (x10 | telets *9/L) tio) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence Listing 1: Sequence (†) AP, Cro | 3.19 Hem Subject Subje | atological Calc. Da cycle and monoc gulation Te Subject hemical la isit Calc. Cycle rCl, Glucos | laborator tte Hem (g ytes. st Visit boratory Date n | Time y value oglobin g/dl) values Total (mg/ | No. of c (125 m) es† Calculate cycle I Bilirubin dl) | wB (x10* | Taken accord | eutrophil<br>x10*9/L) | s Lyr<br>(x<br>epeat | nphocyte (10*9/L) I LT LI U/L) (x | s Pla (x10 | telets *9/L) tio) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence Listing 1: Sequence (†) AP, Cro | 3.19 Hem Subject Derit, RBC 3.20 Coag Subject V Eatinine, C 3.22 Perfe | atological Calc. Da cycle and monoc gulation Te Subject hemical lal isit Calc. Cycle rCl, Glucos | laborator tte Hem (§ ytes. st Visit boratory Date n e, CPK, C | Time y value oglobin y/dl) values Total (mg/ | No. of 6 (125 m) es Calculate cycle I Bilirubin dl) | WB (x10* | Taken accord | eutrophil<br>x10*9/L) Ro | s Lyr<br>(x<br>epeat | nphocyte (10*9/L) I LT LI J/L) (x | s Pla (x10) NR (ra DH ULN) | telets *9/L) tio) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence Listing 1: Sequence (†) AP, Cro | 3.19 Hem Subject Derit, RBC 3.20 Coag Subject V Eatinine, C 3.22 Perfe | atological Calc. Da cycle and monoc gulation Te Subject hemical la isit Calc. Cycle rCl, Glucos | laborator tte Hem (§ ytes. st Visit boratory Date n e, CPK, C | Time y value oglobin g/dl) values Total (mg/ | No. of 6 (125 m) es Calculate cycle I Bilirubin dl) | wB (x10* | Taken accord | eutrophil<br>x10*9/L) | s Lyr<br>(x<br>epeat | nphocyte (10*9/L) I LT LI U/L) (x | s Pla (x10) NR (ra DH ULN) | telets *9/L) tio) |
| Listing 1: Sequence (†) Hemato Listing 1: Sequence Listing 1: Sequence (†) AP, Cro | 3.19 Hem Subject Subje | atological Calc. Da cycle and monoc gulation Te Subject hemical lal isit Calc. Cycle rCl, Glucos | laborator tte Hem (g ytes. St Visit boratory Date n e, CPK, C atus Not | Time y value oglobin y/dl) values Total (mg/ | No. of 6 (125 m) es Calculate cycle I Bilirubin dl) | wB (x10* Direct (mg/d) GGT, To | Taken accord | eutrophil<br>x10*9/L) Ro | s Lyr<br>(x<br>epeat | nphocyte (10*9/L) I LT LI J/L) (x | S Pla (x10) NR (ra DH ULN) C, Mg, | telets *9/L) |

| Sequence | Subject | Not done | Visit | Date | Heart rate | Systolic | Diastolic | Temperature |
|---|---|---|---|---|---|---|---|---|
| | | | | | (bpm) | (mmHG) | (mmHG) | (°C) |
| | 3.25 Electroc | | | | | | | |
| sequence | Subject Visit | Date | | | Specify PR | Heart Q7 | | t's Not done |
| | | | don | e | | | terval correc | |
| | | | | | (ms | ec) (bpm) (m | sec) QT | protocol, specify |
| | | | | | | | | specify |
| | | _ | | | | | | |
| Listing 1. Sequence | 3.26 Concom<br>Subject | | diagnostic j<br>ocedure | Date Date | Indicati | ion AE/N | AU UN | Comments |
| requence | Subject | PI | ocedure | Date | maicau | IOII AE/I | VIII ( | Comments |
| isting 1 | 3.27 LVEF | | | | | | | |
| | | eason Not | t done Vi | sit Date | Method | Value Lowe | r limit Resi | ult Abnorma |
| | | nically | | | | | | specify |
| | ind | licated | | | | | | |
| icting 1 | 3.28 Signs an | d cumpton | ne | | | | | |
| Sequence | | u sympton<br>S&S | | .† Grade | Onset dat | te Still | End date | Related to: |
| requeriee | Buoject | Descri | | . Grade | Onset dat | Ong.at | Ena date | related to. |
| | | | • | | | C1D1? | | |
| †)SOC, N | MedDRA PT | | | | | | | |
| | 3.29 Adverse | events | | | | | | |
| 1 | | | | | | | | |
| sequence | Subject AE. | † G | | _ | _ | elationship A | | |
| | | † G | | Onset Ong.<br>date | End Ong. R | _ | ction Serious<br>ken criteria | |
| | Subject AE. MedDRA PT | † G | | _ | _ | _ | | |
| †)SOC, M | | | | _ | _ | _ | | |
| †)SOC, M<br>Listing 1 | MedDRA PT | nmary | | _ | date eath Life | ta Requires/ | ken criteria | |
| †)SOC, M<br>Listing 1 | MedDRA PT<br>3.30 SAE sun | nmary | | date | date eath Life | Requires/g prolongs | Admissio | ı |
| †)SOC, M<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. | nmary | | date me Start Do | date eath Life | ta Requires/ | Admissio | on Discharge . |
| †)SOC, M<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT | nmary<br>se AE | † Outco | me Start Do | eath Life<br>threatenin | Requires/ g prolongs hospitalization | Admissio<br>date | n Discharge .<br>date ‡ |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant delayers | nmary<br>se AE | † Outco | me Start Do | eath Life<br>threatenin | Requires/ g prolongs hospitalization | Admissio<br>date | n Discharge .<br>date ‡ |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT | nmary<br>se AE | † Outco | me Start Do | eath Life<br>threatenin | Requires/ g prolongs hospitalization | Admissio<br>date | n Discharge .<br>date ‡ |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant delayers | nmary<br>se AE<br>lisability/inve, nullifica | † Outco | me Start Do | eath Life<br>threatenin | Requires/ g prolongs hospitalization | Admissio<br>date | n Discharge .<br>date * |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persistengent trans | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati | nmary se AE lisability/incove, nullifications | † Outco | me Start Dodate me Start Dodate ngenital anor | eath Life threatenin maly, other med | Requires/ g prolongs hospitalization dically importa | Admissio<br>date<br>on | n Discharge .<br>date * |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persistengent trans<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi | nmary se AE lisability/incove, nullifications | † Outco | me Start Do<br>date | eath Life<br>threatenin | Requires/<br>g prolongs<br>hospitalization | Admissio<br>date<br>on | on Discharge . date ‡ vent, infectious |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persistengent trans | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi | nmary se AE lisability/incove, nullifications | † Outco | me Start Dodate me Start Dodate ngenital anor | eath Life threatenin maly, other med | Requires/ g prolongs hospitalization dically importa | Admissio<br>date<br>on | on Discharge . date ‡ vent, infectious |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>gent trans<br>Listing 1<br>Sequence<br>†)ATC1, | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi | nmary se AE disability/inve, nullification | capacity, containing reason cation | me Start Dodate me Start Dodate ngenital anor | eath Life threatenin maly, other med | Requires/ g prolongs hospitalization dically importa | Admissio<br>date<br>on | on Discharge . date ‡ vent, infectious |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>gent trans<br>Listing 1<br>Sequence<br>†)ATC1, | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos | nmary se AE disability/inve, nullification | capacity, containing reason cation | me Start Dodate me Start Dodate ngenital anor | eath Life threatenin maly, other med | Requires/ g prolongs hospitalization dically importa | Admissio<br>date<br>on | on Discharge . date ‡ vent, infectious |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persistengent transl<br>Listing 1<br>Sequence<br>†)ATC1, | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos | nmary se AE disability/inve, nullification | † Outco | me Start Do date ngenital anor Dose Free (units) | eath Life threatenin naly, other med | Requires/<br>g prolongs<br>hospitalization<br>dically important | Admissio date on ant serious ev | on Discharge . date * vent, infectious on AE/MH |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>igent trans<br>Listing 1<br>Sequence<br>†)ATC1,<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos | nmary se AE disability/inve, nullification | † Outco | me Start Do date ngenital anor Dose Free (units) | eath Life threatenin naly, other med | Requires/<br>g prolongs<br>hospitalization<br>dically important | Admissio date on ant serious ev | on Discharge . date * vent, infectious on AE/MH |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>gent trans<br>Listing 1<br>Sequence<br>†)ATC1,<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos: 3.33 Pharmac | nmary se AE lisability/inve, nullification tic procedu | capacity, contained reason cation Route | me Start Do date ngenital anor Dose Free (units) | eath Life threatenin maly, other med uency Start date Date | Requires/ g prolongs hospitalization dically importate End Ongoinate Result | Admissio date on ant serious ev | on Discharge . date ‡ vent, infectious on AE/MH Comments |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>gent trans<br>Listing 1<br>Sequence<br>†)ATC1,<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos | nmary se AE lisability/inve, nullification tic procedu | capacity, contation reason cation Route ures/Tests Subject | me Start Dodate me Start Dodate ngenital anor Dose Frec (units) Test | eath Life threatenin maly, other med uency Start date Date | Requires/ g prolongs hospitalization dically importate End Ongoinate Result | Admissio date on ant serious even untserious e | on Discharge date ** vent, infectious on AE/MH Comments |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>gent trans<br>Listing 1<br>Sequence<br>†)ATC1,<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos: 3.33 Pharmac | nmary se AE lisability/inve, nullification tic procedu | capacity, contation reason cation Route ures/Tests Subject | me Start Do date ngenital anor Dose Free (units) | eath Life threatenin maly, other med uency Start date Date | Requires/ g prolongs hospitalization dically importate End Ongoinate Result | Admissio date on ant serious ev | on Discharge . date * vent, infectious on AE/MH Comments |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persiste<br>gent trans<br>Listing 1<br>Sequence<br>†)ATC1,<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos: 3.33 Pharmac | nmary se AE lisability/inve, nullification tic procedu | capacity, contation reason cation Route ures/Tests Subject | me Start Dodate me Start Dodate ngenital anor Dose Frec (units) Test | eath Life threatenin maly, other med uency Start date Date | Requires/ g prolongs hospitalization dically importate End Ongoinate Result | Admissio date on ant serious even untserious e | on Discharge date ** vent, infectious on AE/MH Comments |
| †)SOC, M<br>Listing 1<br>Sequence<br>†)SOC, M<br>‡)Persistengent transformation of the<br>disting 1<br>Sequence<br>†)ATC1,<br>Listing 1<br>Sequence | MedDRA PT 3.30 SAE sun Subject Cas id. MedDRA PT ent/significant d smitted, narrati 3.31 Concom Subject Medi ATC4 3.32 Diagnos: 3.33 Pharmac | nmary se AE disability/ineve, nullification tic procedutic p | capacity, contain reason cation Route ures/Tests Subject umple Samp | me Start Do date Dose Free (units) Test le Samp. De window | eath Life threatenin maly, other med uency Start date Date | Requires/ g prolongs hospitalization dically importate End Ongoinate Result | Admissio date on ant serious even untserious e | on Discharge date ** vent, infectious on AE/MH Comments |

Listing 13.35 Alpha-1-acid glycoprotein and Interleukin 6

| Sequence | Subject | Visit | Sample taken | Date | Comments |
|---|---|---|---|---|---|
| Listing 13.36 | End of treatment | | | | |
| Sequence | Subject | Primary Reaso | on End of Treatment | t Speci | fy |
| Listing 13.37 | Follow up - Furt | her antitumor therap | ies | | |
| Sequence | Subject | Antitumor The | rapy description | Star | t date |
| Listing 13.38 | Off study | | | | |
| Sequence | Subject | Off Study Date | Primary reason | Specify | Never treated, |
| | | | | | specify |
| Listing 13.39 | Death report form | n | | | |
| Sequence | Subject | Death date | Cause | Specify | Autopsy? |
| | | | of death | | |
| Listing 13.40 | Investigator com | ments | | | |
| Sequence | Subject | Page name | Instance | Variable | Comments |

# 14 APPENDIX V: BIMO Listings

The following listings will be provided following the recommended standardized formats according to the draft Guidance for Industry Standardized Format for Electronic Submission of NDA and BLA Content for the Planning of Bioresearch Monitoring (BIMO) Inspections for CDER Submissions (February 2018) and the associated Bioresearch Monitoring Technical Conformance Guide Containing Technical Specifications.

https://www.fda.gov/downloads/Drugs/DevelopmentApprovalProcess/FormsSubmissionRequirements/UCM332466.pdf

https://www.fda.gov/downloads/Drugs/DevelopmentApprovalProcess/FormsSubmissionRequirements/UCM332468.pdf

| | 4.1 Site lev | vei summary | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Site | | Patients<br>Screene | | | atients End o<br>Treatment | of Patio | ents Off Study |
| Listing | 14.2 Conse | ented subject | s by site | | | | | |
| Site | Subject | Informed<br>Consent date | Screening failure? | Date of<br>Screening<br>failure | Met<br>Eligibility | | Details Tre | eated Date of First treatment |
| Listing | 14.3 Seque | ence assignm | ent by site | | | | | |
| Site | e | Subject | Trea | atment Sequenc | e | DA Start da | ate Firs | t Intended dose |
| Listing<br>Site | 14.4 Disco | ontinuations b<br>End of tr<br>Reas | eatment I | End of treatmen specify | t, C | off-study<br>date | Off stud<br>Reason | |
| Listing | 14.5 Study | population by | • | | | | | |
| Site | Subject | Enrolled p | opulation 1 | PK population | Rease | on Safe | ety population | n Reason |
| Listing | 14.6 Inclus | sion and excl | usion criteria | by Site | | | | |
| Listing<br>Site | | sion and excl | usion criteria<br>Eligibility req | • | Cr | iterion identi | fier I/E | I/E details |
| Site | Su | | Eligibility req | • | Cr | iterion identi | fier I/E | I/E details |
| Site | Su | rse events by Adverse | Eligibility req | uirements? | Cr<br>Relationship<br>Specify | | fier I/E Seriousness Criteria | |
| Site Listing Site | Subject | rse events by Adverse | Site CI- CTC SAE rade | uirements? Onset End I | Relationship | Action | Seriousness | |

| Listing 14.9 Concomitant medication | |
|---|---|
| Site Subject Medication type Medication Reason Route/Dose(Units)/Time Start End date Indication | cation AE/MH |
| †ATC1, ATC4 | |
| Listing 14.10 Individual Laboratory Measurements by site | |
| Site Subject Cycle Examination Laboratory Hematocrit RBC WBC Neutro (x10*9/L) (x10* | |
| †Lymphocytes, Monocytes, Platelets, INR, AST, ALT, AP, LDH, Creatinine, CrCl, Glucose, CPK, Cl GGT, Total Proteins, Total Bilirubin, Direct Bilirubin, Albumin, CRP, Na, K, Mg, Ca. | PK-MB fraction, |
| Listings 14.11 Electrocardiogram by Site | |
| | azett's Not done orrected within T protocol, specify |
| Listings 14.12 LVEF by Site | |
| Site Subject Visit Date Not Done Method LVEF (%) Range Abnormality Sp. Lower Limit | pecify Reason<br>for<br>Clinically<br>Indicated<br>Repeat |

# 15 APPENDIX VI: ICH Listings

In accordance with the International Conference on Harmonization (ICH) E-3 guideline, patient listings specified as section 16.2 will be prepared.

| Listing 16.2.1 Discontinued Patient | ts |
|-------------------------------------|----|
|-------------------------------------|----|

| Cubicat | Institution | Trantad | Cycles | First infusion | Last infusion | Reason for end | Comments |
|---|---|---|---|---|---|---|---|
| Subject | Institution | Treated | received | date | date | of treatment | Comments |

#### Listing 16.2.2 Protocol Deviations

| Subject Deviation type Description | |
|------------------------------------|----------------|
| Subject Deviation type Description | Deviation type |

#### Listing 16.2.3 Patients excluded from the efficacy analysis

Not applicable

#### Listing 16.2.4 Demographic data

| Subject | Tumor | Stage <sup>†</sup> | Λαο | Gender | Race | ECOG | Weight | Height | BSA | Prior | Prior | Prior |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | type | Stage | Age | Gender | Race | ECOG | (kg) | (cm) | $(m^2)$ | radiotherapy | surgery | agents |
| †At diagn | ocic | | | | | | | | | | | |

<sup>†</sup>At diagnosis

Listing 16.2.5 Compliance and/or drug concentration data

| | Lurbinect | edin | | | | | | | Bosentan | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | First<br>Intended<br>dose<br>(mg/m²) | Start<br>date<br>(First<br>cycle) | Start<br>date<br>(Second<br>cycle) | Total<br>dose<br>(mg/m²) | Dose intensity (mg/m²/ wk) | Relative dose intensity (%) | Delays† | Reductions <sup>†</sup> | Taken by protocol | Reason |

<sup>†</sup>Delays/reductions will be nested for each patient (cycle and reason of delay/reduction), e.g. C2 hematological toxicity

#### Listing 16.2.6 Individual efficacy response data

Not applicable

#### Listing 16.2.7 Adverse Event listing (each patient)

| Cubicat | Adverse | SOC PT | Grade | CAE | Onset | End | | Action | Seriousness | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Event | SOC PI | Grade | SAE | date | date | Relationship | taken | criteria | |

#### Listing 16.2.8 Individual Laboratory Measurements by Patient

| | | | Hematocrit | RBC | WBC<br>(x10*9/L) | Neutrophils (x10*9/L) | † |
|---|---|---|---|---|---|---|---|
| Subject | Cycle | Examination date Laboratory | Std. value | Std. value | Std. value | Std. value | Std. value |

<sup>†</sup>Lymphocytes, Monocytes, Platelets, INR, AST, ALT, AP, LDH, Creatinine, CrCl, Glucose, CPK, CPK-MB fraction, GGT, Total Proteins, Total Bilirubin, Direct Bilirubin, Albumin, CRP, Na, K, Mg, Ca.

#### 16 APPENDIX VI: VERSION HISTORY

# 16.1 History of Changes

Minor clarifications/modifications have been added to the SAP v1.0 date on 17 February 2021 during the programing tasks.

A brief summary is include below:

- In order to maintain the consistency in safety analysis groups (Sequence 1 vs Sequence 2 and lurbinectedin administered in combination vs lurbinectedin alone) some table's titles has been clarified and updated.
- Some listings/variables from Appendix IV: DB Listings have been deleted for containing duplicate information.
- Some minor comments for clarification have been added. Minor corrections will not be described below.

Detailed changes are presented in the next pages. Changes are highlighted in *Italic bold* and text removed has been <del>crossed out</del>.

#### APPENDIX I (PATIENTS DISPOSITION)

#### 10.1.1 Patients Disposition

Listing 10.1.1.4 Non-evaluable patients

| Not Evaluable for | Sequence | Subject | Reason(s) |
|-------------------|----------|---------|-----------|
| Safety | | | |
| PK | | | |

#### 10.2.1 Demographic and Other Baseline Characteristics

Table 10.2.1.1 Baseline characteristics: Adequate contraception

| _ | S1 (TR) | | S2 ( | (RT) | To | tal |
|---|---------|---|------|------|----|-----|
| | N | % | N | % | N | % |

Adequate contraception

Yes

No

NA (For Male)

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

## 10.2.5 Physical Examination, ECOG, Vital Signs, LVEF and ECG

Table 10.2.5.6 Baseline characteristics: ECG<sup>†</sup> pre infusion

| S1 ( | TR) | S2 ( | RT) | То | otal |
|------|-----|------|-----|----|------|
| N | % | N | % | N | % |

Result

Normal

Abnormal

Significant abnormalities

Non-significant abnormalities

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable.

† Worst result of the three ECGs replicates will be used as a baseline value.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 10.2.5.10 Baseline characteristics: LVEF

| S1 (TI | R) | | S2 (RT | ) | | Total | |
|--------|----|---|--------|---|---|-------|---|
| <br>N | % | 1 | | % | N | | % |

Result

Normal

Abnormal

Significant abnormalities

Non-significant abnormalities

Notes: Percentage is based on number of patients by total and sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

### APPENDIX II (SAFETY ANALYSIS)

#### 11.2.1 Display of Adverse Events

Table 11.2.1.2 **Treatment** Related<sup>†</sup> (or with unknown relationship) Adverse Events. Worst grade per patient treatment

| | | BOS+-LUR | <del>rbi</del><br>L <b>rb</b> | L | RB alone | |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| SOC/F1 | N % | N % | N % | N % | N % | N % |

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable.

BOS, bosentan; LRB, lurbinectedin.

Table 11.2.1.3 Lurbinectedin related<sup>†</sup> Adverse Events. Worst grade per patient treatment

| | | BOS+-LU | RBI<br>LRB | Ł | <del>URBI</del> LRB | alone |
|---|---|---|---|---|---|---|
| SOC/PT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| SOC/P1 | N % | N % | N % | N % | N % | N % |

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

† Related to lurbinectedin or with unknown relationship

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship

Table 11.2.1.4 Bosentan related Adverse Events. Worst grade per patient treatment

BOS+ **LURBI alone LURB HLRB** All grades  $Gr \ge 3$  $Gr \ge 4$ All grades  $Gr \ge 3$ SOC/PT % Ν % Ν N % N 9/0

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

Table 11.2.1.5 Related<sup>†</sup> (or with unknown relationship) Adverse Events. Worst grade per eyele patient

| | tal | Total | | S2 (RT) | | | (TR) | S1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| N % N | ≥ 3 Gr ≥ 4 | | | $Gr \ge 3$ | | $Gr \ge 4$ | ≥ 3 | Gr | | | SOC/PT |
| | % N % | % N % | N % N % | N % | N % | N % | % | N | % | N | · |

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable

Table 11.2.1.6 Lurbinectedin related<sup>†</sup> Adverse Events. Worst grade per cycle

| | | | S1 | (TR) | | | | , | <del>S2 (</del> R | <del>T)</del> | | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <del>SOC/PT</del> | A<br>gra | | Gr | <del>≥ 3</del> | Gr | <del>≥ 4</del> | A<br>gra | | Gr | <del>≥ 3</del> | Gr | <del>≥ 4</del> | oro | <del>des</del> | Gr | <u>≥ 3</u> | Gr | <del>≥ 4</del> |
| | N | % | N | % | N | <del>%</del> | N | % | N | <del>%</del> | Ŋ | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients by total and sequence, when applicable.

Table 11.2.1.7 Bosentan related† Adverse Events. Worst grade per cycle

| | | | <u>S1</u> | <del>(TR)</del> | | | | _ | S2 ( | <del>RT)</del> | | | | | | <del>Total</del> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <del>SOC/PT</del> | A<br>gra | | Gr | <del>≥ 3</del> | Gr | <u>≥4</u> | A<br>gra | <del>.ll</del><br><del>des</del> | Gr | <del>≥ 3</del> | Gr | <u>≥4</u> | oro | <del>des</del> | Gr | <u>≥ 3</u> | Gr | <del>≥</del> 4 |
| | N | <del>%</del> | N | % | N | <del>%</del> | N | <del>%</del> | N | <del>%</del> | N | % | N | % | N | <del>%</del> | N | % |

Notes: Percentage is based on number of patients by total and sequence, when applicable.

<sup>†</sup> Related to bosentan or with unknown relationship BOS, bosentan; LRB, lurbinectedin.

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†-</sup>Related to lurbinectedin or with unknown relationship

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

<sup>†</sup> Related to bosentan or with unknown relationship

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.2.1.86 Adverse Events regardless of relationship. Worst grade per patient treatment

| | | | BOS+<br><del>LURB</del><br><del>I</del> LRB | LURBI LRB alone |
|---|---|---|---|---|
| SOC/DT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades $Gr \ge 3$ $Gr \ge 4$ |
| SOC/PT | N % | N % | N % | N % N % N % |

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

BOS, bosentan; LRB, lurbinectedin.

Table 11.2.1.9-8Adverse Events regardless of relationship. Worst grade per eyele patient

| | | | S1 | (TR) | | | | | S2 | (RT) | | | | | 7 | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | A<br>gra | | Gr | ≥ 3 | Gr | ≥4 | | ll<br>des | Gr | ≥ 3 | Gr | ≥4 | | ll<br>des | Gr | ≥ 3 | Gr | ≥ 4 |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients by total and sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 11.3.1 Serious Adverse Events

Table 11.3.1.1 **Treatment** Related<sup>†</sup> (or with unknown relationship) SAEs. Worst grade per patient treatment

| SOC/PT $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | | | BOS+<br><del>LURB</del><br><del>I</del> LRB | LURBI LRB alone |
|---|---|---|---|---|
| N % N % N % N % N % N % | COC/DT | All grades | $Gr \ge 3$ $Gr \ge 4$ | All grades $Gr \ge 3$ $Gr \ge 4$ |
| | SOC/P1 | N % | N % N % | N % N % N % |

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

Table 11.3.1.2 Lurbinectedin related† SAEs. Worst grade per patient treatment

| | | - | BOS+<br><del>LURBI</del><br>L <b>RB</b> | <del>LURBI</del> LR | B alone |
|---|---|---|---|---|---|
| SOC/PT | All grades | Gr ≥ 3 | $Gr \ge 4$ | All grades $Gr \ge 3$ | $Gr \ge 4$ |
| SOC/F1 | N % | N % | N % | N % N % | N % |

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship BOS, bosentan; LRB, lurbinectedin.

<sup>†</sup> Related to lurbinectedin or with unknown relationship

Table 11.3.1.3 Bosentan related† SAEs. Worst grade per patient treatment

| | | BOS+ <del>LUR</del> | <del>Bi</del><br>L <b>rb</b> | LURBI LRB alone |
|---|---|---|---|---|
| SOC/DT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades $Gr \ge 3$ $Gr \ge 4$ |
| SOC/P1 | N % | N % | N % | N % —N % —N % |

. . .

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable

BOS, bosentan; LRB, lurbinectedin.

Table 11.3.1.4 **Treatment** Related† (or with unknown relationship) SAEs. Worst grade per eyele patient

| | | | S1 | (TR) | | | | | S2 | ' ( | ) | | | | Tota | 1 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | | dl<br>des | Gr | ≥ 3 | Gr | ≥4 | A<br>gra | des | Gr | ≥ 3 | Gr | ≥4 | A<br>gra | des | Gr | ≥ 3 | Gr | ≥4 |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

. . .

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test

Table 11.3.1.5 Lurbinectedin related \* SAEs. Worst grade per cycle

| | | | S1 | (TR) | | | | | | (RT | ) | | | | Total | ļ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | A<br>gra | | Gr | <u>≥ 3</u> | Gr | | A<br>gra | H<br><del>des</del> | Gr | <u>≥ 3</u> | Gr | ≥4 | A<br>gra | doc | Gr | <u>≥ 3</u> | Gr | <u>≥4</u> |
| | N | <del>%</del> | N | <del>%</del> | N | <del>%</del> | N | <del>%</del> | N | <del>%</del> | N | <del>%</del> | N | <u>0/</u> | N | <del>%</del> | N | % |

. . .

Notes: Percentage is based on number of patients by total and sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.3.1.6 Bosentan related<sup>†</sup> SAEs. Worst grade per cycle

| | | | (111) | | | | | | (RT) | <del>)</del> | | | - | <del>Total</del> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT g | All<br>rades | Gr: | ≥3 | Gr : | ≥4 | A<br>grad | | Gr | <u>≥3</u> | Gr | ≥4 | A<br>gra | | Gr | <u>≥3</u> | Gr | <u>~</u> -4 |
| 4 | <del>%</del> | N | % | N | % | Ŋ | <del>%</del> | N | % | N | <del>%</del> | Ŋ | % | N | % | N | % |

•••

Notes: Percentage is based on number of patients by total and sequence, when applicable.

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.3.1.75 SAEs regardless of relationship. Worst grade per patient treatment

| | | | BOS+<br><del>LURB</del><br><b>ILRB</b> | | LRB <del>LU</del> | RBI alone |
|---|---|---|---|---|---|---|
| COC/DT | All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ | $Gr \ge 4$ |
| SOC/PT | N % | N % | N % | N % | N % | N % |

• •

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

<sup>†</sup> Related to bosentan or with unknown relationship

<sup>†</sup> Related to both or lurbinectedin or bosentan or with unknown relationship

<sup>†</sup>Related to lurbinectedin or with unknown relationship

<sup>†</sup> Related to bosentan or with unknown relationship

Table 11.3.1.86 SAEs regardless of relationship. Worst grade per eyele patient

| | | | S1 | (TR) | | | | | S2 | (RT | ) | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC/PT | A<br>gra | | Gr | ≥ 3 | Gr | ≥4 | A<br>gra | ll<br>des | Gr | ≥ 3 | Gr | ≥4 | | .ll<br>des | Gr | ≥ 3 | Gr | ≥4 |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

. . .

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

# 11.4.1 Hematological Abnormalities

Table 11.4.1.1 Hematological abnormalities: Worst grade per patient treatment

| | | BOS+<br><del>LURB</del><br><del>I</del> LRB | | LURBI LRB alone |
|---|---|---|---|---|
| All grades | $Gr \ge 3$ | $Gr \ge 4$ | All grades | $Gr \ge 3$ $Gr \ge 4$ |
| N % | N % | N % | N % | N % N % |

Anemia

Leukopenia

Lymphopenia

Neutropenia

Thrombocytopenia

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

BOS, bosentan; LRB, lurbinectedin.

Table 11.4.1.4 Hematological abnormalities: Worst grade per eyele patient

| | | S1 | (TR) | | | | ( | S2 (R | (T) | | | | | Tot | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| A<br>gra | | Gr | ≥ 3 | Gr | ≥4 | | .ll<br>.des | Gr | ≥ 3 | Gr | ≥4 | | ll<br>des | Gr | ≥ 3 | Gr | ≥4 |
| N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Anemia

Leukopenia

Lymphopenia

Neutropenia

Thrombocytopenia

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 11.4.2 Biochemical Abnormalities

Table 11.4.2.1 Biochemical abnormalities: Worst grade per patient treatment

| | | BOS+<br>LURB<br>ILRB | | | <del>LURBI</del> I | L <b>RB</b> alone |
|---|---|---|---|---|---|---|
| All grades | $Gr \ge 3$ | $Gr \ge 4$ | All gra | ades | $Gr \ge 3$ | $Gr \ge 4$ |
| N % | N % | N % | N | % | N % | N % |

ALT increase AST increase

Notes: Percentage is based on number of patients by total and sequence is based on number of patients by treatment, when applicable

\*Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia, hypocalcemia.

BOS, bosentan; LRB, lurbinectedin.

Table 11.4.2.4 Biochemical abnormalities: Worst grade per eyele patient

| <br>*** | | | | | ~ · B- | | | <i>J</i> | Pere | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | S1 | (TR) | | | | | | RT) | | | | | To | otal | | |
| | des. | Gr | ≥3 | Gr | ≥4 | | All<br>ides | Gr | ≥ 3 | Gr | ≥4 | | ll<br>des | Gr | ≥ 3 | Gr | ≥4 |
| N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

ALT increase

AST increase

Notes: Percentage is based on number of patients by total and sequence is based on number of patients in total and by sequence, when applicable.

Notes: Percentage is based on number of patients by total and sequence, when applicable.

\*Creatinine increased, hyperglycemia, hypoglycemia, CPK increased, GGT increased, bilirubin increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia, hypocalcemia

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

#### 11.4.3 Laboratory Values Over Treatment

Table 11.4.3.2 Time course for neutrophils and platelets

| | <del>\$1 (TF</del> | <del>2)</del> BOS+LRB | —————————————————————————————————————— | AT)LRB<br>alone | | Total |
|---|---|---|---|---|---|---|
| | N | Median<br>(range) | N | Median<br>(range) | N | Median<br>(range) |
| Neutropenia (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Nadir day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |
| Thrombocytopenia (Grade≥3) | | | | | | |
| Onset day | | | | | | |

Onset day

Nadir day

Recovery day

Days of recovery to grade ≤2

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

Table 11.4.3.4 Time course for AST and ALT

| | S | <del>1 (TR)</del> BOS+LRB | Total | | | |
|---|---|---|---|---|---|---|
| | N | Median<br>(range) | N | Median<br>(range) | N | Median (range) |
| AST (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Peak day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |
| ALT (Grade≥3) | | | | | | |
| Onset day | | | | | | |
| Peak day | | | | | | |
| Recovery day | | | | | | |
| Days of recovery to grade ≤2 | | | | | | |

S1, Sequence 1; S2, Sequence 2; TR, test-reference; RT, reference-test.

BOS, bosentan; LRB, lurbinectedin.

# APPENDIX IV (DB Listings)

| Listing 13.1 | Screening | (I) | Ì |
|--------------|-----------|-----|---|
|--------------|-----------|-----|---|

| Sequence Su | ıbject | Informed | PGt | Planned | Age | Tumor | EC3 I | EC4 | PCR date | PCR result | Eligibility |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | consent | sub-study | initiation | | type | | | | | |

## Listing 13.3 Sponsor Approval Form

| Sequence | <del>Subject</del> | <del>Approval</del> | Comments | <b>Lurbinectedin</b> | <b>Lurbinectedin</b> |
|---|---|---|---|---|---|
| | | | | in combination (mg/m2) | alone (mg/m2) |

## **Listing 13.4 Randomization details**

| Sequence | <del>Subject</del> | Ready to be | Treatment | <del>Treatment</del> | Date/Time |
|---|---|---|---|---|---|
| | | randomized | Sequence | Description | of randomization |

#### Listing 13.53 Study registration/Randomization details

| Sequence | Subject | Registration Date of | Treatment | Treatment | Screening |
|---|---|---|---|---|---|
| | | <b>Randomization</b> Randomization | Sequence | Description | failure date |